Statistical Analysis Plan, Version 5.0 Date Issued: 06-JAN-2025

# ModernaTX, Inc.

#### Protocol mRNA-1083-P101

# A Phase 1/2, Randomized, Observer-blind, Active-Control Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-based Influenza and SARS-CoV-2 Multi-component Vaccines in Healthy Adults

# Statistical Analysis Plan

**SAP Version 5.0** 

**Version Date of SAP: 06-JAN-2025** 

Prepared by:

PPD, part of Thermo Fisher Scientific

929 North Front Street

Wilmington, NC 28401-3331

United States

# TABLE OF CONTENTS

| TABLE OF CONTENTS | 2 |
|--------------------------------------------------------|----|
| LIST OF TABLES | 5 |
| LIST OF FIGURES | |
| LIST OF ABBREVIATIONS | 6 |
| SUMMARY OF MAJOR CHANGES IN SAP VERSION | 8 |
| 1. INTRODUCTION | 9 |
| 2. PART 1 | 10 |
| 2.1. Study Objectives | |
| 2.1.1. Primary Objectives | 10 |
| 2.1.2. Secondary Objectives | 10 |
| 2.1.3. Exploratory Objectives | 10 |
| 2.2. Study Endpoints | |
| 2.2.1. Primary Endpoints | |
| 2.2.2. Secondary Endpoints | 11 |
| 2.2.3. Exploratory Endpoints | 12 |
| 2.3. Study Design | 12 |
| 2.3.1. Overall Study Design | 12 |
| 2.3.2. Statistical Hypotheses | |
| 2.3.3. Sample Size and Power | 15 |
| 2.3.4. Randomization | 15 |
| 2.4. Blinding and Unblinding | 15 |
| 2.5. Analysis Sets | 16 |
| 2.5.1. Randomization Set | |
| 2.5.2. Full Analysis Set (FAS) | |
| 2.5.3. Per Protocol (PP) Set | |
| 2.5.4. Safety Set | |
| 2.5.5. Solicited Safety Set | |
| 2.6. Statistical Analysis | |
| 2.6.1. General Considerations | |
| 2.6.2. Background Characteristics | 23 |
| 2.6.2.1. Participant Disposition | 23 |
| 2.6.2.2. Demographics and Baseline Characteristics | 25 |
| 2.6.2.3. Medical History | 26 |
| 2.6.2.4. Prior and Concomitant Medications | |
| 2.6.2.5. Study Exposure | 27 |
| 2.6.2.6. Major Protocol Deviations | |
| 2.6.2.7. COVID-19 Impact | |
| 2.6.3. Safety Analysis | |
| 2.6.3.1. Solicited Adverse Reactions | |
| 2.6.3.2. Unsolicited Treatment-Emergent Adverse Events | |
| 2.6.3.3. Death | 35 |
| 2.6.3.4. Clinical Safety Laboratory Tests | |
| 2.6.3.5. Vital Signs | |
| 2.6.3.6. Pregnancy Testing | |
| 2.6.3.7. Other Safety Data | 37 |

| 2.6.4. Immunogenicity Analysis | 38 |
|--------------------------------------------------------|----|
| 2.6.4.1. Secondary Immunogenicity Endpoints | 39 |
| 2.6.4.2. Exploratory Immunogenicity Endpoints | |
| 2.6.5. Exploratory Analysis | 45 |
| 2.6.5.1. Efficacy Analysis | 45 |
| 2.6.5.2. Influenza Infection | 45 |
| 2.6.5.3. SARS-CoV-2 Infection | 47 |
| 2.6.6. Other Exploratory Endpoints | 48 |
| 2.6.7. Planned Analyses | |
| 2.6.7.1. Interim Analysis | 49 |
| 2.6.7.2. Final Analysis | 49 |
| 3. PART 2 | |
| 3.1. Study Objectives | 50 |
| 3.1.1. Primary Objectives | |
| 3.1.2. Secondary Objectives | |
| 3.1.3. Exploratory Objectives | |
| 3.2. Study Endpoints | |
| 3.2.1. Primary Endpoints | |
| 3.2.2. Secondary Endpoints | |
| 3.2.3. Exploratory Endpoints | 51 |
| 3.3. Study Design | 52 |
| 3.3.1. Overall Study Design | |
| 3.3.2. Statistical Hypotheses | |
| 3.3.3. Sample Size and Power | |
| 3.3.4. Randomization | 55 |
| 3.4. Blinding and Unblinding | |
| 3.5. Analysis Sets | |
| 3.5.1. Randomization Set | |
| 3.5.2. Full Analysis Set (FAS) | 55 |
| 3.5.3. Per Protocol (PP) Set | |
| 3.5.4. Safety Set | |
| 3.5.5. Solicited Safety Set | 57 |
| 3.6. Statistical Analysis | 57 |
| 3.6.1. General Considerations | |
| 3.6.2. Background Characteristics | |
| 3.6.2.1. Participant Disposition | |
| 3.6.2.2. Demographics and Baseline Characteristics | |
| 3.6.2.3. Medical History | 60 |
| 3.6.2.4. Prior and Concomitant Medications | 60 |
| 3.6.2.5. Study Exposure | |
| 3.6.2.6. Major Protocol Deviations | 60 |
| 3.6.3. Safety Analysis | |
| 3.6.3.1. Solicited Adverse Reactions | |
| 3.6.3.2. Unsolicited Treatment-Emergent Adverse Events | |
| 3.6.3.3. Death | |
| 3.6.3.4. Vital Signs | 62 |

| 3.6.3.5. Pregi | nancy Testing | 62 |
|---|---|---|
| 3.6.3.6. Other | r Safety Data | . 62 |
| 3.6.4. Immun | ogenicity Analysis | . 62 |
| 3.6.4.1. Prima | ary Immunogenicity Endpoints | . 63 |
| 3.6.4.2. Secon | ndary Immunogenicity Endpoints | . 67 |
| 3.6.4.3. Expl | oratory Immunogenicity Endpoints | . 67 |
| 3.6.5. Other I | Exploratory Endpoints | . 68 |
| 3.6.6. Planne | d Analyses | . 68 |
| 3.6.6.1. Interi | m Analysis | . 68 |
| 3.6.6.2. Final | Analysis | . 68 |
| 4. CHANGE | S FROM PLANNED ANALYSIS IN PROTOCOL | . 69 |
| 5. REFERE | NCES | . 70 |
| 6. APPENDI | CES | . 71 |
| Appendix A | Schedule of Activities (SoA) | .71 |
| I. Part 1 | | . 71 |
| II. Part 2 | | . 74 |
| Appendix B | Analysis Visit Windows | |
| Appendix C | Imputation Rules for Missing Prior/Concomitant Medications and Non-Study | |
| Vaccinations | 78 | |
| Appendix D | Imputation Rules for Missing AE dates | |
| Appendix E | Severity Grading of Laboratory Abnormalities | .81 |
| Appendix F | Severity Grading of Vital Sign Abnormalities | . 83 |
| Appendix G | Solicited Adverse Reactions and Grades | . 84 |
| Appendix H | TEAE of Specifical Interest by SMQ | . 86 |

# LIST OF TABLES

| Table 1 Study Arm(s) and Interventions (Part 1) | 13 |
|---|---|
| Table 2 Sample Size Determination (Part 1) | 15 |
| Table 3 Exclusion Condition for Dosing Errors (Part 1) | 17 |
| Table 4 As Treated Grouping Scheme (Part 1) | 18 |
| Table 5 Definition for Subgroups by Cohort A and B (Part 1) | 23 |
| Table 6 Covariates Included in Different ANCOVA Models (Part 1) | 42 |
| Table 7 Exploratory between-group Immunogenicity comparisons (Part 1) | 43 |
| Table 8 Respiratory and Systemic Symptoms for Protocol-defined ILI (Part 1) | 46 |
| Table 9 Study Arm(s) and Interventions (Part 2) | 53 |
| Table 10 Sample Size Determination (Part 2) | 55 |
| Table 11 Exclusion Condition for Dosing Errors (Part 2) | 56 |
| Table 12 As Treated Grouping Scheme (Part 2) | 57 |
| Table 13 Definition for Subgroups (Part 2) | 59 |
| Table 14 Covariates Included in Different ANCOVA Models (Part 2) | 64 |
| Table 15 Between-group Immunogenicity comparisons (Part 2) | 66 |
| Table 16 Analysis Visit Windows for Immunogenicity Assessments | 77 |
| Table 17 Prior, Concomitant, and Post Categorization of a Medication | 79 |
| LIST OF FIGURES | |
| Figure 1 Study Schema (Part 1) | 14 |
| Figure 2 Study Schema (Part 2) | 54 |

# LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|--------------|-------------------------------------------------|
| AE | adverse event |
| AESI | adverse event of special interest |
| ANCOVA | analysis of covariance |
| AR | adverse reaction |
| bAb | binding antibody |
| BMI | body mass index |
| CI | confidence interval |
| CDC | US Centers for Disease Control and Prevention |
| CMQ | Customized MedDRA Query |
| COVID-19 | coronavirus disease 2019 |
| CRO | contract research organization |
| CSP | clinical study protocol |
| CSP | clinical study protocol clinical study report |
| DHHS | Department of Health and Human Services |
| DSMB | |
| | Data Safety Monitoring Board |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EDC . | electronic data capture |
| eDiary | electronic diary |
| EoS | end of study |
| FAS | Full Analysis Set |
| FSH | follicle-stimulating hormone |
| GLSM | geometric least square mean |
| GM | geometric mean |
| GMFR | geometric mean fold rise |
| GMR | geometric mean ratio |
| GMT | geometric mean titer |
| HA | hemagglutinin |
| HAI | hemagglutination inhibition |
| IA | Interim analysis |
| ILI | influenza-like illness |
| IM | intramuscular |
| IP | investigational product |
| IRT | interactive response technology |
| LLOQ | lower limit of quantification |
| MAAE | medically attended adverse event |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mRNA | messenger ribonucleic acid |
| nAb | neutralizing antibody |
| NP | nasopharyngeal |
| PP | Per-Protocol |
| PsVNA | pseudovirus neutralization assay |
| PT | preferred term |
| RT-PCR | reverse transcriptase polymerase chain reaction |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SARS-CoV-2 | severe acute respiratory syndrome coronavirus 2 |
| SAS | Statistical Analysis System |
| SCR | seroconversion rate |
| SD | standard deviation |

| Abbreviation | Definition |
|--------------|-------------------------------------------|
| SMQ | Standardized MedDRA Query |
| SOC | system organ class |
| SoA | schedule of activities |
| SRR | seroresponse rate |
| TEAE | treatment-emergent adverse event |
| ULOQ | upper limit of quantification |
| WHO | World Health Organization |
| WHODD | World Health Organization drug dictionary |


# SUMMARY OF MAJOR CHANGES IN SAP VERSION

| SAP<br>Version | Section # and Name | Description of Change |
|---|---|---|
| V2.0 | 5.3 Per Protocol (PP) Set | Clarified existing language for conditions/medications that affect the immune response. |
| V2.0 | 6.1 General Considerations | Clarified that all subgroups are based on eCRF entries unless otherwise stated. Added definition for Baseline SARS-CoV-2 Status and added this Baseline SARS-CoV-2 Status to Table 5, as a subgrouping factor to be used in table summaries. |
| V2.0 | 6.2.2 Demographics and Baseline Characteristics | Added 3 categorical baseline variables: Baseline SARS-CoV-2 RT-PCR Results, Elecsys Anti-SARS-CoV-2 Results, and Baseline SARS-CoV-2 Status. |
| V2.0 | 6.3.2 Unsolicited Treatment-<br>Emergent Adverse Events | Updated to reflect only Solicited ARs that meet SAE criteria are recorded on the Reactogenicity eCRF. |
| V2.0 | 6.4.2 Immunogenicity Analysis | Updated wording in 6.4.2.2 Analytical summaries, and added a new Table 6 to clarify the covariates used in the ANCOVA analyses. Renumbered later tables and added clarifying language to Table 7. Removed bar-plot of ANCOVA-based GMT. |
| V3.0 | 6.2.4 Prior and Concomitant<br>Medications | "Antipyretic or analgesic medication within 28 days postinjection" item removed |
| V3.0 | 6.4.2.1. Analysis of Secondary<br>Immunogenicity Endpoints | For GMFR, values below LLOQ imputed to LLOQ |
| V3.0 | 6.4.2.2 Analytical summaries | Added D181 GMT/GMR; added figure for D181 GMFR, SCR, SRR, and GMR |
| V3.0 | 6.5.1.2 SARS-CoV-2 Infection | Asymptomatic SARS CoV 2 infection language removed |
| V3.0 | Appendix H TEAE of Specifical Interest by SMQ | SMQ table updated |
| V4.0 | Global update | Part 2 added to the SAP per protocol amendment 1 dated 16-<br>Jan-2024 and protocol amendment 2 dated 14 Mar 2024 |
| V5.0 | 3.6.4.1. Primary<br>Immunogenicity Endpoints | Updated the "Covariate(s)" column in Table 14, by adding "Log-transformed baseline antibody value" for all rows. |

#### 1. Introduction

This statistical analysis plan (SAP), which describes the planned analyses for Study mRNA-1083-P101, is based on the most recent approved clinical study protocol amendment (CSP), dated 14-MAR-2024, and the most recent approved electronic case report form (eCRF), dated 31-MAY-2024.

In addition to the principal features of analyses for this study described in Section 9 of the protocol, this SAP provides statistical analysis details/data derivations. It also documents modifications or additions to the analysis plan that are not "principal" in nature and result from information that was not available at the time of protocol finalization.

Study mRNA-1083-P101 is a phase 1/2, randomized, observer-blind, active-control study to evaluate the safety, reactogenicity, and immunogenicity of mRNA-based Influenza and SARS-CoV-2 multi-component vaccines in healthy adults.

The study is divided into 2 parts: Part 1 and Part 2. Part 1 (Phase 1/2) includes adults who are 18 to <80 years and Part 2 (Phase 2 Extension) includes adults who are 18 to <50 years.

Approximately 1744 participants will be enrolled in the overall clinical trial.

PPD Biostatistics and Programming team, designee of Moderna Biostatistics and Programming department, will perform the statistical analysis of the safety, reactogenicity, and immunogenicity data; Statistical Analysis System (SAS) Version 9.4 or higher will be used to generate all statistical outputs (tables, figures, listings, and datasets). The SAP will be finalized and approved prior to the primary analysis clinical database lock and treatment unblinding for the study. If the methods in this SAP differ from the methods described in the protocol, the SAP will prevail.

In this document, study vaccination, intervention administration, injection of investigational product (IP)/investigational vaccine, dosing, and injection are used interchangeably. Treatment group, investigational treatment arm, vaccination group are used interchangeably.

#### 2. Part 1

# 2.1. Study Objectives

#### 2.1.1. Primary Objectives

The primary objective is to evaluate the safety and reactogenicity of study intervention administration across study treatment arms.

## 2.1.2. Secondary Objectives

The secondary objectives are:

- To evaluate the humoral immune responses to vaccine-matched strains for influenza and SARS-CoV-2 across study treatment arms at Day 29
- To evaluate the humoral immune responses to vaccine-matched strains for influenza and SARS-CoV-2 across study treatment arms at all evaluable humoral immunogenicity time points

## 2.1.3. Exploratory Objectives

The following exploratory objectives may be assessed:

- To evaluate the humoral immune responses to vaccine-mismatched strains for influenza and SARS-CoV-2 across study treatment arms
- To evaluate the humoral immune responses against vaccine-matched and vaccinemismatched strains for influenza and SARS-CoV-2 across study treatment arms
- To evaluate the cellular immune responses against influenza and SARS-CoV-2 in a subset of participants
- To further characterize the immune response to influenza and SARS-CoV-2 across study treatment arms
- To assess the occurrence of clinical influenza and COVID-19 in study participants and characterize their immune response to infection and viral isolates

#### 2.2. Study Endpoints

# 2.2.1. Primary Endpoints

The primary objective will be evaluated by the following endpoints:

- Solicited local and systemic adverse reactions (ARs) through 7 days after injection
- Unsolicited AEs through 28 days after injection
- Unsolicited severe adverse events through 28 days after injection
- Unsolicited medically attended adverse events (MAAEs) from Day 1 to Day 181/End of Study (EoS)
- Unsolicited adverse events of special interest (AESIs) from Day 1 to Day 181/EoS
- Serious adverse events (SAEs) from Day 1 to Day 181/EoS
- Unsolicited AEs leading to discontinuation from Day 1 to Day 181/EoS

#### 2.2.2. Secondary Endpoints

The secondary objective will be evaluated by the following endpoints:

- Geometric mean titer (GMT) and geometric mean fold rise (GMFR) at Day 29 compared with Day 1 by hemagglutination inhibition (HAI) assay for influenza and by pseudovirus neutralization assay (PsVNA) for SARS-CoV-2
- Influenza: Percentage of participants with seroconversion, defined as a Day 29 titer CCI if Baseline is CCI or a 4-fold or greater rise if Baseline is CCI in anti-HA antibodies measured by HAI assay
- SARS-CoV-2: Percentage of participants with seroresponse, defined as a Day 29 titer
   ≥4-fold if Baseline is ≥LLOQ or ≥4 × LLOQ if Baseline titer is <LLOQ in
   neutralizing antibody (nAb) titers measured by PsVNA</li>
- GMT and GMFR at all evaluable timepoints compared with Day 1 by HAI for influenza and PsVNA for SARS-CoV-2
- Influenza: Percentage of participants with seroconversion at all evaluable timepoints
- SARS-CoV-2: Percentage of participants with seroresponse at all evaluable timepoints

#### 2.2.3. Exploratory Endpoints

The exploratory objectives may be evaluated by the following endpoints:

- GMT and GMFR at all evaluable timepoints compared with Day 1 by HAI for influenza and PsVNA for SARS-CoV-2
- Influenza: Percentage of participants with seroconversion to vaccine mismatched strains at all evaluable timepoints
- SARS-CoV-2: Percentage of participants with seroresponse to vaccine mismatched strains at all evaluable timepoints
- GMT and GMFR at all evaluable timepoints compared with Day 1 by alternative methods, including, but not limited to: microneutralization assay for influenza or ligand-binding assay for SARS-CoV-2
- Frequency, magnitude, and phenotype of virus-specific T-cell and B-cell responses measured by flow cytometry or other methods
- Perform targeted repertoire analysis of B-cells and T-cells after vaccination
- Frequency, specificities, or other endpoints to be determined for the further characterization of immune responses
- Frequency of RT-PCR-confirmed clinical influenza and COVID-19
- Assessment of immune responses to infection and viral isolates

#### 2.3. Study Design

#### 2.3.1. Overall Study Design

**Part 1** of the study is a Phase 1/2 randomized, stratified, observer-blind, active-control study to evaluate the safety, reactogenicity, and immunogenicity of mRNA-1083 compositions and dose levels compared with active-control vaccines mRNA-1010, mRNA-1283.222, mRNA-1273.222, and licensed active-control vaccines, Fluarix<sup>®</sup> and Fluzone<sup>®</sup> HD (Cohort A only) in healthy adults  $\geq$ 18 to <80 years of age (Cohort A is in adults  $\geq$ 65 to <80 years of age and Cohort B is in adults  $\geq$ 18 to <65 years of age).

Approximately 1224 participants will be enrolled into 1 of 2 age cohorts: Cohort A for adults  $\geq$ 65 to <80 years of age or Cohort B for adults  $\geq$ 18 to <65 year of age. In Cohort A,

approximately 600 participants will be randomized (in equal allocation ratio) into the investigational treatment arms, stratified by influenza vaccine status in the most recent influenza season (received or not received since September 2022). In Cohort B, approximately 624 participants will be randomized (in equal allocation ratio) into the investigational treatment arms, stratified by 2 age groups:  $\geq 18$  to <50 years and  $\geq 50$  to <65 years of age and by influenza vaccine status in the most recent influenza season (received or not received since September 2022). Approximately 50% of the participants in Cohort B will be  $\geq 50$  to <65 years of age. Table 1 lists the details of study cohorts and dose levels for study vaccine administration. All participants will receive a single intramuscular (IM) injection of study intervention administered in a deltoid muscle on Day 1.

Table 1 Study Arm(s) and Interventions (Part 1)

| Cohort A Arms:<br>(≥65 to <80<br>years),<br>n=50/arm, 600 | Cohort B Arms:<br>(≥18 to <65<br>years),<br>n=52/arm, 624 | Intervention | Total mRNA Dose (μg) | Intervention<br>Type |
|---|---|---|---|---|
| total | total | | | |
| NA | B1 | mRNA-1083.1 | CCI | IP |
| A2 | B2 | mRNA-1083.1 | | IP |
| A3 | В3 | mRNA-1083.1 | | IP |
| A4 | B4 | mRNA-1083.2 | | IP |
| A5 | B5 | mRNA-1083.2 | | IP |
| A6 | В6 | mRNA-1083.2 | | IP |
| A7 | В7 | mRNA-1083.3 | | IP |
| A8 | В8 | mRNA-1010. | | Non-IP experimental comparator |
| A9 | В9 | mRNA-<br>1283.222 | | Non-IP experimental comparator |
| A10 | B10 | mRNA-<br>1273.222 | | Non-IP experimental comparator |
| A11 | B11 | mRNA-1010 | | Non-IP experimental comparator |
| A12 | B12 | Fluarix | | Licensed vaccine comparator |
| A13 | NA | Fluzone HD | | Licensed vaccine comparator |

Abbreviations: HD=high dose; IP=investigational product; mRNA=messenger ribonucleic acid; NA=not applicable; SARS-Cov-2=severe acute respiratory syndrome coronavirus 2.

Total mRNA dose is rounded to the nearest μg

All participants of the study will participate in a Screening period (up to 28 days before Day 1), treatment period (single dose of vaccine on Day 1), and a follow-up period (up to 6 months after


vaccination). The study schema is presented in Figure 1. Please refer to the Schedule of Activities (SoA) available in Appendix A.

Figure 1 Study Schema (Part 1)



Abbreviations: HD=high dose; mRNA=messenger ribonucleic acid

# 2.3.2. Statistical Hypotheses

This clinical trial does not have formal statistical hypothesis testing planned for the primary objective (safety and reactogenicity). The total sample sizes planned are considered sufficient to provide descriptive summary of the safety and reactogenicity across study treatment arms within each age Cohort for respective parts.

#### 2.3.3. Sample Size and Power

The sample size for this study is not driven by statistical assumptions for formal hypothesis testing. Approximately 1224 participants will be enrolled at an evenly allocated ratio across the 12 treatment arms in Cohort A for adults ≥65 to <80 years of age and 12 treatment arms in Cohort B for adults ≥18 to <65 years of aged, with 50 participants planned for each arm in Cohort A (600 participants in total) and 52 participants planned for each arm in Cohort B (624 participants in total) (Table 2). Approximately 50 participants in each group receiving an investigational injection have approximately 87% (or 92%) probability to observe at least 1 participant with an AE given the true underlying incidence rate of AE is 4% (or 5%).

**Table 2 Sample Size Determination (Part 1)** 

| Sample Size | True AE Rate | Probability of 0 AEs | Power to Detect at Least 1 AE |
|---|---|---|---|
| 50 | 2.0% | 36.4% | 63.6% |
| 50 | 3.0% | 21.8% | 78.2% |
| 50 | 4.0% | 13.0% | 87.0% |
| 50 | 5.0% | 7.7% | 92.3% |

Abbreviation: AE = adverse event.

#### 2.3.4. Randomization

Randomization will be performed using an interactive response technology (IRT) by a 3<sup>rd</sup> party vendor.

- In Cohort A, approximately 600 participants will be randomized (in equal allocation ratio) into the investigational treatment arms, stratified by influenza vaccine status in the most recent influenza season (received or not received since September 2022).
- In Cohort B, approximately 624 participants will be randomized (in equal allocation ratio) into the investigational treatment arms, stratified by 2 age groups: ≥18 to <50 years and ≥50 to <65 years of age and by influenza vaccine status in the most recent influenza season (received or not received since September 2022). Approximately 50% of the participants in Cohort B will be ≥50 to <65 years of age.</p>

#### 2.4. Blinding and Unblinding

The planned analyses including a potential Day 8 interim analysis and the Day 29 interim analysis are described in Section 2.6.7 of this SAP. For further details on preidentified sponsor

and CRO team members (identified by role), and the level of unblinding (treatment group level unblinding and/or subject level unblinding) at the IAs and the Final analysis, please refer to the study Data Blinding Plan.

## 2.5. Analysis Sets

#### 2.5.1. Randomization Set

The randomization set consists of all participants who are randomly assigned. Participants will be included in the vaccination group to which they are randomized.

#### 2.5.2. Full Analysis Set (FAS)

The FAS consists of all participants who are randomly assigned and receive the study intervention. Participants will be analyzed according to the group to which they were randomized.

### 2.5.3. Per Protocol (PP) Set

The PP Set in Part 1 consists of all participants in the FAS who comply with the injection schedule, comply with the timings of immunogenicity blood sampling to have a Baseline and at least 1 post-injection assessment at Day 29 (-7 to +14 days), have no documented infection (confirmed by RT-PCR test) of either influenza or SARS-CoV-2 on Day 1 and up to Day 29 (Day 29 immunogenicity assessment + 7 days), have no major dosing error, and have no major protocol deviations or conditions/medications that affect the immune response. The PP Set will be used as the primary analysis set for analyses of immunogenicity in Cohort A or B unless otherwise specified. Participants will be analyzed according to the group to which they were randomized.

The major dosing error ranges, available in Table 3, will be used to determine participant exclusion from the PP analysis populations:

**Table 3 Exclusion Condition for Dosing Errors (Part 1)** 

| Randomized Group | <b>Exclusion Conditions</b> |
|---|---|
| mRNA-1083.1 ( μg) | Any of the following received:<br>mRNA-1083.1 ≤ μg OR mRNA-1083.1 > μg OR<br>mRNA-1083.2 OR mRNA-1083.3 OR |
| | mRNA-1010 OR mRNA-1010. OR mRNA-1283.222 OR mRNA-1273.222 OR Fluarix OR Fluzone HD |
| mRNA-1083.1 ( μg) | Any of the following received:<br>mRNA-1083.1 ≤ CCI μg OR mRNA-1083.1 > CCI μg OR |
| | mRNA-1083.2 OR mRNA-1083.3 OR<br>mRNA-1010 OR mRNA-1010. OR mRNA-1283.222 OR mRNA-1273.222 |
| | OR Fluarix OR Fluzone HD |
| mRNA-1083.1 ( μg) | Any of the following received:<br>mRNA-1083.1 ≤ μg OR mRNA-1083.1 > μg OR<br>mRNA-1083.2 OR mRNA-1083.3 OR |
| | mRNA-1010 OR mRNA-1010. OR mRNA-1283.222 OR mRNA-1273.222 |
| mRNA-1083.2 (CCI μg) | OR Fluarix OR Fluzone HD Any of the following received: |
| mκινΑ-1065.2 ( <b>Δ61</b> μg) | mRNA-1083.2 <b>CCI</b> μg OR mRNA-1083.2 > <b>CCI</b> μg OR mRNA-1083.1 OR mRNA-1083.3 OR |
| | mRNA-1010 OR mRNA-1010 OR mRNA-1283.222 OR mRNA-1273.222 OR Fluarix OR Fluzone HD |
| mRNA-1083.2 ( μg) | Any of the following received: |
| | mRNA-1083.2 $\leq$ CCI $\mu$ g OR mRNA-1083.2 $>$ CCI $\mu$ g OR |
| | mRNA-1083.1 OR mRNA-1083.3 OR |
| | mRNA-1010 OR mRNA-1010. OR mRNA-1283.222 OR mRNA-1273.222 OR Fluzix OR Fluzone HD |
| mRNA-1083.2 ( μg) | Any of the following received: |
| ( | mRNA-1083.2 ≤ CCI μg OR mRNA-1083.2 > CCI μg OR mRNA-1083.1 OR mRNA-1083.3 OR |
| | mRNA-1010 OR mRNA-1010. OR mRNA-1283.222 OR mRNA-1273.222 OR Fluarix OR Fluzone HD |
| mRNA-1083.3 (CCI μg) | Any of the following received:<br>mRNA-1083.3 ≤ CCI μg OR mRNA-1083.3 > CCI μg OR |
| | mRNA-1083.1 OR mRNA-1083.2 OR |
| | mRNA-1010 OR mRNA-1010 OR mRNA-1283.222 OR mRNA-1273.222 OR Fluarix OR Fluzone HD |
| mRNA-1010. (μg) | Any of the following received: |
| <del>-</del> - | mRNA-1010. 4 ≤ 1 μg OR mRNA-1010. 5 > 1 μg OR |
| | mRNA-1083.1 OR mRNA-1083.2 OR mRNA-1083.3 OR |
| | mRNA-1010 OR mRNA-1283.222 OR mRNA-1273.222 OR Fluarix OR |
| mRNA-1283.222 (μg) | Fluzone HD Any of the following received: |
| μg) | mRNA-1283.222 $\leq$ µg OR mRNA-1283.222 $>$ µg OR |
| | mRNA-1083.1 OR mRNA-1083.2 OR mRNA-1083.3 OR |
| | mRNA-1010 OR mRNA-1010. OR mRNA-1273.222 OR Fluarix OR |
| | Fluzone HD |
| mRNA-1273.222 ( μg) | Any of the following received: |
| | mRNA-1273.222 ≤ |
| | mRNA-1083.1 OR mRNA-1083.2 OR mRNA-1083.3 OR |
| | mRNA-1010 OR mRNA-1010 OR mRNA-1283.222 OR Fluarix OR Fluzone HD |
| mRNA-1010 ( μg) | Any of the following received: |
| · | mRNA-1010 ≤ µg OR mRNA-1010 > OR |

| Randomized Group | <b>Exclusion Conditions</b> |
|------------------|-----------------------------------------------------------|
| | mRNA-1083.1 OR mRNA-1083.2 OR mRNA-1083.3 OR |
| | mRNA-1010 OR mRNA-1283.222 OR mRNA-1273.222 OR Fluarix OR |
| | Fluzone HD |
| Fluarix | Any of the following received: |
| | Fluarix ≤ 30 μg OR |
| | mRNA-1083.1 OR mRNA-1083.2 OR mRNA-1083.3 OR |
| | mRNA-1010 OR mRNA-1010. OR mRNA-1283.222 OR mRNA-1273.222 |
| | OR Fluzone HD |
| Fluzone HD | Any of the following received: |
| | Fluzone HD ≤ 120 μg OR |
| | mRNA-1083.1 OR mRNA-1083.2 OR mRNA-1083.3 OR |
| | mRNA-1010 OR mRNA-1010. OR mRNA-1283.222 OR mRNA-1273.222 |
| | OR Fluarix |

Note: " $\leq x.x \mu g$ " includes the missing injection (i.e. 0.0  $\mu g$ ) of the planned vaccination.

# 2.5.4. Safety Set

The Safety Set consists of all participants who are randomly assigned and receive the study intervention. The Safety Set will be used for all analyses of safety, except for the solicited ARs. Participants will be included in the vaccination group corresponding to what they actually received according to the as treated scheme given below in Table 4.

**Table 4 As Treated Grouping Scheme (Part 1)** 

| Group Name | Inclusion condition |
|---|---|
| mRNA-1083.1 (CCI μg) | Any dose of mRNA-1083.1 $\leq$ CCl $\mu$ g |
| mRNA-1083.1 (CCI μg) | Any dose of mRNA-1083.1 $>$ CCl $\mu g$ and $\leq$ $\mu g$ |
| mRNA-1083.1 (CCI μg) | Any dose of mRNA-1083.1 $>$ $\frac{\cos \mu}{\mu}$ and $\leq$ $\frac{\cos \mu}{\mu}$ |
| mRNA-1083.2 (CCI μg) | Any dose of mRNA-1083.2 ≤ CCI μg |
| mRNA-1083.2 ( <sup>CCI</sup> μg) | Any dose of mRNA-1083.2 $>$ CCI $\mu$ g and $\leq$ CCI $\mu$ g |
| mRNA-1083.2 (CCI μg) | Any dose of mRNA-1083.2 > CCl μg |
| mRNA-1083.3 (CCI μg) | Any dose of mRNA-1083.3 |
| mRNA-1010. (CCI μg) | Any dose of mRNA-1010. |
| mRNA-1283.222 (CCI μg) | Any dose of mRNA-1283.222 |
| mRNA-1273.222 ( <sup>CCI</sup> μg) | Any dose of mRNA-1273.222 |
| mRNA-1010 ( μg) | Any dose of mRNA-1010 |
| Fluarix | Any dose of Fluarix |
| Fluzone HD | Any dose of Fluzone HD |

#### 2.5.5. Solicited Safety Set

The solicited safety set consists of all participants in the safety set who contribute any solicited AR data. The solicited safety set will be used for the analyses of solicited ARs and participants will be included in the vaccination group corresponding to what they actually received (as treated).

#### 2.6. Statistical Analysis

The SoA is provided in the Appendix A.

#### 2.6.1. General Considerations

All analyses will be conducted using SAS Version 9.4 or higher. Statistical outputs (tables, figures, listings, and datasets) will refer study participants as participants and will use injection of IP and injection interchangeably.

Continuous variables will be summarized using the following descriptive summary statistics: the number of participants (n), mean, standard deviation (SD), median, Q1 and Q3 (only for summaries specified below), as well as minimum (min), and maximum (max). For the summary statistics of all numerical variables unless otherwise specified, the display precision will follow programming standards.

Summaries that require Q1 and Q3 for descriptive statistics:

- Demographic and baseline characteristics
- Study duration
- Characteristics of solicited adverse reactions within 7 days after injection
- Descriptive summaries of antibody levels

Categorical variables will be summarized using counts and percentages. When count data are presented, the percentage will be suppressed when the count is zero in order to draw attention to the non-zero counts. A row denoted "Missing" will be included in count tabulations where specified on the shells to account for dropouts and missing values. The denominator for all percentages will be the number of participants in the treatment group within the analysis set of interest, unless otherwise specified.

**Baseline value**, unless specified otherwise, is defined as the most recent non-missing measurement (scheduled or unscheduled) collected before the dose/time of IP in this study. For immunogenicity tests and nasal swab tests, the baseline is defined as the most recent non-missing result/measurement (scheduled or unscheduled) collected before or on the date of injection (Day 1). If there are multiple valid results on the same date, the largest value will be considered in the immunogenicity baseline derivation.

**Baseline SARS-CoV-2 status** is determined by using virologic and serologic evidence of SARS-CoV-2 infection on or before Day 1.

- Positive SARS-CoV-2 status at Baseline is defined as a positive RT-PCR test for SARS-CoV-2, and/or a positive serology test based on bAb specific to SARS-CoV-2 nucleocapsid on or before Day 1.
- Negative status at Baseline is defined as a negative RT-PCR test for SARS-CoV-2 and a negative serology test based on bAb specific to SARS-CoV-2 nucleocapsid on or before Day 1.

# The following analysis periods of safety analyses will be used:

- Throughout the Study: from the day of vaccination (Day 1) and continues through the earliest date of (study completion, discontinuation from the study, or death).
- Within 7 days after injection: this period includes the day of vaccination and 6 subsequent days, or up to the study discontinuation or death, whichever comes earlier.
   This analysis period will be used for solicited local and systemic AR that occur during this time.
- Up to 28 days after injection: starts from the day of vaccination (Day 1) and spans 28 days to include the day of vaccination and 27 subsequent days, or up to the study discontinuation or death, whichever comes earlier. This analysis period will be used as the primary analysis period for safety analyses including unsolicited AE, except for solicited AR, unless specified otherwise.

#### **Study day relative to the injection** will be calculated as below:

- a) study day prior to the injection will be calculated as: date of assessment/event date of the injection (resulting in negative study day);
- b) study day on or after the date of the injection will be calculated as: date of assessment/event date of the injection + 1;

**Duration of an event** will be calculated as (Event end date – Event start date +1). The duration of the study will be calculated for the participants included in the safety set:

• Since randomization: date of last visit (as recorded on End of Study [EoS] eCRF) – date of randomization + 1,

• Since study injection: date of last visit (as recorded on End of Study [EoS] eCRF) – date of injection + 1.

If the last visit date on the EoS eCRF page is missing, then the latest of either the cut-off date or the last available visit date will be employed. The durations of solicited ARs will be calculated as: reaction end date – reaction start date +1, regardless of whether the AR is intermittent or continued or if the solicited AR continues beyond 7 days.

**For calculation regarding antibody levels/titers**, antibody values reported as below the lower limit of quantification (LLOQ) will be replaced by  $0.5 \times \text{LLOQ}$ . Values that are greater than the upper limit of quantification (ULOQ) will be converted to the ULOQ if actual values are not available. Missing results will not be imputed.

**Unscheduled visits:** Unscheduled visit measurements will be included in the analyses as follows:

- In scheduled visit windows per specified visit windowing rules (Appendix B).
- In the derivation of baseline/last on-treatment measurements.
- In the derivation of maximum/minimum on-treatment values and maximum/minimum change from baseline values for safety analyses.
- In individual Participant data listings.

**Visit window rules:** The analysis visit windows for protocol-defined visits are provided in Appendix B.

#### **Incomplete/missing data:**

- Imputation rules for missing prior/concomitant medications, non-study vaccinations and procedures are provided in Appendix C.
- Imputation rules for missing AE dates are provided in Appendix D.
- Other incomplete/missing data will not be imputed, unless specified otherwise.

**Table layouts** will be presented according to vaccination group. First for the overall participants, then by subgroups as given in Table 5.

For Part 1, all the statistical analyses will be performed and presented by Cohort A and Cohort B, separately. The following vaccination groups will be used for summary purposes for Cohort A and for Cohort B tables and figures outputs, respectively:

#### Cohort A:

- Fluarix
- Fluzone HD
- mRNA-1010 μg
- mRNA-1010. μg
- mRNA-1273.222 μg
- mRNA-1283.222 μg
- mRNA-1083.1 <sup>CCI</sup> μg
- mRNA-1083.1 <sup>CCI</sup> μg
- mRNA-1083.2 CCI μg
- mRNA-1083.2 <sup>CCI</sup> μg
- mRNA-1083.2 μg
- mRNA-1083.3 CCI μg
- All mRNA-1083.1 (all mRNA-1083.1 vaccination groups combined; applicable to safety and reactogenicity analyses only)
- All mRNA-1083.2 (all mRNA-1083.2 vaccination groups combined; applicable to safety and reactogenicity analyses only)
- Overall (All vaccination groups combined; details are available below)

#### Cohort B:

- Fluarix
- mRNA-1010 cc μg
- mRNA-1010. μg
- mRNA-1273.222 μg
- mRNA-1283.222 ccl μg
- mRNA-1083.1 cc μg
- mRNA-1083.1 <sup>CCI</sup> μg

- mRNA-1083.1 cc μg
- mRNA-1083.2 CCI μg
- mRNA-1083.2 ccl μg
- mRNA-1083.2 μg
- mRNA-1083.3 CCI μg
- All mRNA-1083.1 (all mRNA-1083.1 vaccination groups combined; applicable to safety and reactogenicity analyses only)
- All mRNA-1083.2 (all mRNA-1083.2 vaccination groups combined; applicable to safety and reactogenicity analyses only)
- Overall (All vaccination groups combined; details are available below)

The "Overall" combined group will be presented for baseline summaries such as participant disposition, demographic summaries, concordance of randomization stratum, etc. as well as major protocol deviation, medical history, concomitant medication and study duration summaries.

**Subgroups by Cohort A and B**: For Part 1, the following subgroups will be used for summary purposes, where indicated in this SAP. Unless otherwise specified, all subgroups are based on eCRF.

**Table 5 Definition for Subgroups by Cohort A and B (Part 1)** 

| Cohort Applicable | Subgroup Variable | Categories |
|---|---|---|
| Cohort B only | Age Group | ≥18 to <50 years |
| | | $\geq$ 50 to <65 years |
| Cohort A and B | Influenza vaccine status since | Received previous season flu vaccine |
| | Sept 2022 | Did not receive previous season flu vaccine |
| Cohort A and B | Prior bivalent Covid vaccine | Received prior bivalent Covid vaccine |
| | status | Did not receive prior bivalent Covid vaccine |
| Cohort A and B | Baseline SARS-CoV-2 Status | Positive |
| | | Negative |

#### 2.6.2. Background Characteristics

#### 2.6.2.1. Participant Disposition

The number and percentage of participants in each of the following disposition categories will be summarized by treatment group (as defined in Section 2.6.1) based on the Randomization Set:

- Randomized
- Received study injection
- Completed study
- Prematurely discontinued the study and the reason for discontinuation

This study treatment only consists of a 1-dose, thus discontinuation from study treatment is not applicable to this study. A Participant is considered to have completed the study if he or she has completed the study including the last Day 181 scheduled procedure (SoA).

A Participant disposition listing will be provided, including informed consent, participants who received study injection, participants who completed study, participants who discontinued from study, with reasons for discontinuation.

In addition, randomized participants with any inclusion and exclusion criteria deviation will also be provided in a listing.

The number of participants in the following categories will be summarized based on Participants Screened:

- Number of participants screened
- Number and percentage of screen failure participants and the reason for screen failure

The percentage of participants who screen failed will be based on the number of participants screened. The reason for screen failure will be based on the number of participants who screen failed. A screen failure listing will be provided including information on the screen failed participants and the reasons for screen failure.

The number and percentage of participants in the following Analysis Sets (see Section 0) will be summarized by treatment group (as defined in Section 2.6.1) based on the Randomization Set:

- Randomization Set
- FAS
- PP Set
- Safety Set
- Solicited Safety Set


For Solicited Safety Set, the percentage will be based on the number of participants in the treatment group within the Safety Set (as treated). A summary of reasons for participants excluded from PP will also be provided.

A Randomization listing will be provided including randomization information such as randomization date, number, planned and actual treatment group and stratification used.

An additional listing, including information related to the different Analysis Sets of the randomized participants as well as the reason for exclusion from analysis set will be added.

A separate summary table will include the number and percentage of randomized participants by vaccination group with respect to each combined stratification factor at randomization by IRT (i.e. >18 to <50 years and Received, >18 to <50 years and Not Received,  $\geq$ 50 to <65 years and Received,  $\geq$ 50 to <65 years and Not Received) and by each of the two stratification factors at randomization separately (>18 to <50 vs.  $\geq$ 50 to <65 years; Received vs. Not received).

If IRT and eCRF stratum are not concordant, then a concordance table will be presented, by vaccination group based on the Randomization Set, with the number and percentage of patients in IRT randomization stratum and actual stratum derived from eCRF.

#### 2.6.2.2. Demographics and Baseline Characteristics

Descriptive statistics will be calculated for the following continuous demographic and baseline characteristics:

- Age (years)
- Weight (kg)
- Height (cm)
- Body mass index (BMI) (kg/m<sup>2</sup>)

The number and percentage of participants will be provided for the following categorical variables:

- Age group (≥ 18 to <50 years old, ≥ 50 to < 65 years old for Cohort B, ≥ 65 to <80 years old for Cohort A, separately) per age reported on the eCRF</li>
- Sex (Male, Female)

- Race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, Multiracial, Other, Not Reported, Unknown)
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino, Not Reported, Unknown)
- Influenza vaccine status in the most recent influenza season (received or not received since Sept 2022) per eCRF
- Prior bivalent Covid vaccine status (received or not received) per eCRF
- Childbearing Potential for female participants (Yes/No) and reason if "No"
- Baseline SARS-CoV-2 RT-PCR Results (positive, negative, or missing)
- Baseline Elecsys Anti-SARS-CoV2 Results (positive, negative, or missing)
- Baseline SARS-CoV-2 Status (positive, negative, or missing)

The summaries will be provided separately for all analysis sets (except Randomization Set and Solicited Safety Set) defined in the Section 0. The number and percentage of participants randomized by country and site will be provided as well.

# 2.6.2.3. Medical History

Medical history data will be coded by system organ class (SOC) and preferred term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA).

The number and percentage of participants with any medical history will be summarized by SOC and PT based on the Safety Set. A participant will be counted only once for multiple events within each SOC and PT. SOC will be displayed in internationally agreed order. PT will be displayed in descending order of frequency of the "Overall" group and then alphabetically within SOC.

Medical history data will be presented in a listing.

#### 2.6.2.4. Prior and Concomitant Medications

Prior and concomitant medications and non-study vaccination will be coded using the World Health Organization (WHO) drug dictionary (WHODD). The summary of concomitant medications will be based on the Safety Set. Categorization of prior, concomitant, and post medications and imputation rules for missing/partial dates is summarized in Appendix C.

An overall summary with the number and percentage of participants using concomitant medications and non-study vaccination that continued or newly received at or after the injection, during the 7-day follow-up period (i.e., on the day of injection and the 6 subsequent days) and during the 28 day follow-up period after the injection (i.e., on the day of injection and the 27 subsequent days) will be provided by vaccination group (as defined in Section 2.6.1) as follows:

- Any concomitant medications and non-study vaccination within 7 days postinjection
- Any concomitant medications and non-study vaccination within 28 days post-injection
- Any seasonal influenza or COVID-19 vaccine within 28 days post-injection

An additional summary table of concomitant medications and non-study vaccination that continued or newly received at or after the injection through 28 days will be provided by PT in descending frequency based on "Overall" group.

Medications taken to prevent or treat pain or fever will be collected in the electronic diary (eDiary). A summary table will be provided based on the Solicited Safety Set by vaccination group (as defined in Section 2.6.1), including within 7 days after injection, beyond 7 days after injection, and any time after injection.

Prior, concomitant and post medications and non-study vaccination will be presented in a listing. Medications taken to prevent or treat pain or fever will be presented as well (see Section 2.6.3.1 on solicited ARs listings).

Concomitant Procedures will be presented in a listing.

# 2.6.2.5. Study Exposure

Study vaccine administration data will be presented in a listing. Participants with any dosing errors will also be presented in a separate listing.

Study duration (the study duration calculation is available in Section 2.6.1) will be summarized since randomization, and since the study injection based on Safety Set.

#### 2.6.2.6. Major Protocol Deviations

Major protocol deviations are a subset of protocol deviations that may significantly impact the completeness, accuracy, or reliability of the study data or that may significantly affect a

participant's rights, safety, or well-being. Major protocol deviations rules will be developed and finalized before database lock.

The number and percentage of the participants with each major protocol deviation type will be provided by treatment group (as defined in Section 2.6.1), based on the Randomization Set.

Selected major protocol deviations might impact critical or key study data such as the immune response. Participants with such deviations will be excluded from the PP set. Such major protocol deviations will be determined and documented by Sponsor prior to database lock and unblinding. Reasons of exclusion from PP set will be summarized (see section 2.6.2.1).

Major protocol deviations will be presented in a listing.

#### 2.6.2.7. COVID-19 Impact

A listing will be provided for COVID-19 impact on missed or out of window visits or assessments for participants in Safety Set.

## 2.6.3. Safety Analysis

Safety and reactogenicity will be assessed by clinical review of all relevant parameters, including solicited ARs (local and systemic events), unsolicited AEs, SAEs, AESIs, MAAEs, severe AEs, and AEs leading to withdrawal from study participation.

All safety analyses will be provided by treatment group available in the Section 2.6.1. Participants will be included in the treatment group corresponding to what they actually received and will be based on the Safety Set, except summaries of solicited ARs, which will be based on the Solicited Safety Set unless otherwise specified. Imputation rules for missing/partial dates is detailed in Appendix D.

#### 2.6.3.1. Solicited Adverse Reactions

Solicited ARs are predefined local (at the injection site) and systemic events/symptoms that participants are specifically asked, and which are noted by the participant in their eDiary. The eDiary will solicit daily participant reporting of ARs using a structured checklist from the day of vaccination (Day 1) and for the 6 days after the day of dosing (through Day 7). Solicited ARs include selected signs and symptoms that are typically associated with vaccine reactogenicity.

Local ARs are expected after intramuscular study intervention administration. These are typically mild, transient, and self-limited and may include pain, erythema (redness), swelling/induration (hardness) at the injection site and/or ipsilateral underarm swelling/tenderness. Systemic ARs may also occur after study intervention administration, the majority of which are of mild to moderate in severity. Systemic ARs reported with other mRNA vaccines may include fatigue, headache, myalgia, fever, chills, arthralgia, vomiting and/or nausea.

Reactogenicity refers to the occurrence and intensity of local and systemic ARs commonly following vaccination. Severity grading of reactogenicity will occur automatically based on participant entry into the eDiary according to the grading scales presented in Appendix G modified from the Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials (DHHS, 2007). All solicited ARs (local and systemic) will be considered causally related to dosing.

Any solicited AR that meets any of the following criteria must be entered into the participant's source document and must also be recorded in the participant's Reactogenicity eCRF:

- Solicited local or systemic AR that results in a visit to a healthcare professional (MAAE)
- Solicited local or systemic AR leading to the participant withdrawing from the clinical trial or the participant being withdrawn from the clinical trial by the Investigator (AE leading to withdrawal)
- Solicited local or systemic AR lasting beyond 7 days post-injection
- Solicited local or systemic AR that otherwise meets the definition of an SAE

#### Additionally:

- If a participant reported a solicited AR during the solicited period and did not record the event in the eDiary, the event should be recorded on the Reactogenicity page of the eCRF.
- If the event starts during the solicited period, but continues beyond 7 days after dosing, the participant should notify the site to provide an end date to close out the event on the Reactogenicity page of the eCRF.

• If the participant reported an event after the solicited period (i.e., after Day 7), it should be recorded as an AE on the AE page of the eCRF.

When summarizing the number and percentage of participants with an event, participants will be presented according to the highest severity/toxicity in the summaries by severity/toxicity.

#### 2.6.3.1.1 Overview of Solicited ARs

An overall summary of solicited ARs up to 7 days after study injection (with a toxicity grade of Grade 1 or greater) including the number and percentage of participants, along with the number of events, by vaccination group (as defined in Section 2.6.1) will be presented.

The number and percentage of subjects experiencing any solicited local ARs and solicited systemic ARs of Grade 3 or higher will be provided.

# 2.6.3.1.2 Solicited ARs by Toxicity Grade

An summary of solicited ARs up to 7 days after study injection (with a toxicity grade of Grade 1 or greater) by toxicity grade, including the number and percentage of participants, by vaccination group (as defined in Section 2.6.1) who experience the following will be presented:

- Any solicited ARs,
- Any solicited systemic AR,
- Any solicited local AR,
- Each individual solicited systemic and local AR,

A 2-sided 95% exact CI using the Clopper-Pearson method will also be provided for the percentage of participants with any solicited AR (overall and local, systemic). An additional description for Grade 3 or Above (Grade >=3) will be provided for all above categories.

A summary figure will be produced for local and systemic event rates by toxicity grade.

# 2.6.3.1.3 Solicited ARs by Onset Day

An summary of solicited ARs up to 7 days after study injection (with a toxicity grade of Grade 1 or greater) by onset day (from Day 1 through Day 7), including the number and percentage of

participants, by vaccination group (as defined in Section 2.6.1) who experience the following will be presented:

- Any solicited ARs,
- Any solicited systemic AR,
- Any solicited local AR,
- Each individual solicited systemic and local AR,

The onset of individual solicited AR is defined as the time point after injection (Section 2.6.1) at which the respective solicited AR first occurred.

#### 2.6.3.1.4 Characteristics of Solicited ARs

A descriptive summary of the day of onset and the duration of solicited ARs up to 7 days after study injection (with a toxicity grade of Grade 1 or greater), by vaccination group (as defined in Section 2.6.1) who experience the following will be presented:

- Any solicited ARs,
- Any solicited systemic AR,
- Any solicited local AR,
- Each individual solicited systemic and local AR

The onset of individual solicited AR is defined as the time point after injection (Section 2.6.1) at which the respective solicited AR first occurred. The duration calculation method is available in the Section 2.6.1 as well.

#### 2.6.3.1.5 Other solicited ARs summaries

A summary of solicited ARs persisting beyond 7 days after study injection (with a toxicity grade of Grade 1 or greater) by grades, including the number and percentage of participants, by vaccination group (as defined in Section 2.6.1) who experience the following will be presented:

- Any solicited ARs,
- Any solicited systemic AR,
- Any solicited local AR,
- Each individual solicited systemic and local AR.

Solicited local and systemic ARs (with a toxicity grade of Grade 1 or greater) will be provided in listings. Medications taken to prevent or treat pain or fever will also be presented. All solicited ARs that continue beyond 7 days post-injection (with a toxicity grade of Grade 1 or greater) will be listed as well.

# 2.6.3.2. Unsolicited Treatment-Emergent Adverse Events

A treatment-emergent AE (TEAE) is defined as any event occurring during the study not present before exposure to IP or any event already present that worsens in intensity or frequency after exposure to IP.

An unsolicited TEAE is any AE reported by the participant that is not specified as a solicited AR in the protocol or is specified as a solicited AR but starts outside the protocol-defined period for reporting solicited ARs (i.e., 7 days after study vaccine administration). For analysis and reporting purposes, unsolicited TEAEs will include the following:

- TEAEs that are reported by participants and recorded on the AE eCRF
- Solicited ARs that meet SAE criteria after injection are recorded on the Reactogenicity eCRF

Unsolicited AEs include serious (SAE) and nonserious AEs. Worsening of a pre-existing condition after vaccination will be reported as a new AE.

A MAAE is an AE that leads to an unscheduled visit to a healthcare professional (HCP). This would include visits to a study site for unscheduled assessments (e.g., rash assessment, abnormal laboratory follow-up) and visits to HCPs external to the study site. An AESI is an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program for which ongoing monitoring and immediate notification by the Investigator to the Sponsor is required and documentation is in the form of a case narrative. Such events may require further investigation to characterize and understand them.

All unsolicited AEs reported or observed during the clinical trial will be collected from start of study intervention through 28 days after injection. All AEs leading to study discontinuation, MAAE, SAEs, and AESIs will be collected from the start of study intervention administration until through EoS or discontinuation from the clinical trial.

Unsolicited AEs will be coded according to Medical Dictionary for Regulatory Activities (MedDRA) version 26.0 or higher and presented by MedDRA system organ class (SOC) and preferred term (PT).

Analyses of unsolicited TEAEs will be provided (1) for up to 28 days after vaccination and (2) until EoS visit unless otherwise specified (as defined in Section 2.6.1). SOC will be displayed in an internationally agreed order. PT will be displayed in descending order of frequency of the combined:

• 1083.2 treatment group (mRNA-1083.2 CCI μg, mRNA-1083.2 μg, and mRNA-1083.2 μg), and then alphabetically within each SOC.

When summarizing the number and percentage of participants with an event, participants with multiple occurrences of the same AE or a continuing AE will be counted once. Only the maximum severity level will be presented in the severity/toxicity summaries, and the strongest relationship level will be presented in the relationship summaries.

For the by-severity summaries, the toxicity grade of a solicited AR meeting SAE criteria will be mapped to a severity level of Mild/Grade 1, Moderate/Grade 2, or Severe/ $\geq$  Grade 3, and the maximum severity level in the case of multiple events will be presented.

The following listings containing individual participant AEs data will be provided:

- Any unsolicited AEs,
- Any treatment-related unsolicited AEs,
- Unsolicited serious AEs,
- Unsolicited serious treatment-related AEs,
- Unsolicited severe AEs
- Unsolicited AEs leading to discontinued from the study,
- Unsolicited MAAEs,
- Unsolicited AESIs,

Treatment-emergent AEs will be flagged in all data listings.

In addition, number of participants with occurrences of selected TEAEs of clinical interests identified by SMQ will be summarized up to 28 days after injection and throughout the study.

SMQ will be summarized by PT, if applicable. Detailed description of SMQ is presented in Appendix H. A listing of unsolicited AEs by SMQ will be provided.

#### 2.6.3.2.1 Overview of Unsolicited TEAEs

An overall summary of unsolicited TEAEs, including the number and percentage of participants, by vaccination group (as defined in Section 2.6.1) who experience the following will be presented:

- Any unsolicited AEs,
- Any unsolicited serious AEs,
- Any unsolicited AESI,
- Any unsolicited AEs that are medically attended,
- Any unsolicited AEs leading to study discontinuation,
- Any unsolicited severe (/≥ grade 3) AEs,
- Any unsolicited AEs that are fatal.

The table will also include number and percentage of participants with unsolicited TEAEs that are treatment-related in each of the above categories.

## 2.6.3.2.2 TEAEs by System Organ Class and Preferred Term

The following summary tables of TEAEs will be provided by SOC and PT using frequency counts and percentages (i.e., number and percentage of participants with an event) and number of events by vaccination group (as defined in Section 2.6.1):

- All unsolicited AEs,
- All unsolicited AEs that are treatment-related,
- All unsolicited serious AEs,
- All unsolicited serious AEs that are treatment-related,
- All unsolicited AESI,
- All unsolicited AESI that are treatment-related,
- All unsolicited AEs that are medically attended,
- All unsolicited AEs that are medically attended that are treatment-related,
- All unsolicited severe (grade  $\geq$  3) AEs,

- All unsolicited severe (grade  $\geq$  3) AEs that are treatment-related,
- All unsolicited AEs leading to study discontinuation,

#### 2.6.3.2.3 TEAEs by Preferred Term

Tables of all unsolicited TEAEs will be provided by PT sorted in a descending order starting with the frequency of the combined 1083.2 group (mRNA-1083.2  $\mu$ g, mRNA-1083.2  $\mu$ g, and mRNA-1083.2  $\mu$ g).

#### 2.6.3.2.4 TEAEs by Severity

The following summary tables of TEAEs will be provided by SOC, PT and the maximum severity or toxicity grade using frequency counts and percentages:

- All unsolicited AEs
- All unsolicited AEs that are treatment-related

Summary tables will also be provided by SOC and PT for unsolicited TEAEs that are treatment-related in each of the above categories.

#### 2.6.3.3. Death

Total number of deaths due to any cause and time of death from injection (numeric and by time point window) will be summarized in a table. In addition, number of participants with occurrences of Unsolicited TEAE Leading to Death will be summarized by SOC and PT using frequency counts and percentages. A listing of deaths including cause of death, and a listing of unsolicited AEs in participants who died will be provided.

#### 2.6.3.4. Clinical Safety Laboratory Tests

Safety laboratory tests will consist of white blood cell count, hemoglobin, hematocrit, platelets, AST, ALT, creatinine, alkaline phosphatase, and total bilirubin will be assessed at Screening and Day 8. The Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials (DHHS, 2007) available in Appendix E will be used to categorize clinical laboratory test results.

Observed values and changes from baseline to post-baseline visit (at Day 8) for continuous hematology and serum chemistry parameters will be summarized by vaccination group. A toxicity grade shift table of the hematology and chemistry parameters from baseline to post-baseline visit will be provided as well.

Listing containing individual participant clinical laboratory tests measurements data will be provided for hematology and serum chemistry. Additionally, participant with any abnormal post-baseline laboratory tests measurements where toxicity grade (Grade 2 or higher) will be listed separately: if a participant has a laboratory result with Grade 2 or higher abnormality after injection visit, then all results for that participant will be presented in the listing. The values that are outside the reference ranges will be flagged in a data listing.

If multiple values are collected within a post-baseline visit/timepoint, the last assessment will be used in the by-visit summary tables. Unscheduled visits (including early termination) will not be summarized in by-visit summaries of data but may contribute to either baseline or post-baseline worst-case (maximum, minimum, etc.) values when applicable. All values will be listed.

#### **2.6.3.5. Vital Signs**

Vital sign measurements will include systolic and diastolic blood pressure, heart rate, respiratory rate, and body temperature (preferred route is oral) and will be assessed at Screening and Day 1. On the day of study intervention administration, vital sign measurements will be collected once before and at least 60 minutes after study intervention. Vital signs may be collected at other study visits in conjunction with a symptom-directed physical examination.

Following injection, any abnormal vital sign measurement should be assessed by the Investigator to determine if it meets AE reporting criteria per protocol and reported as an AE in EDC, if appropriate.

The Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical (DHHS, 2007) available in Appendix F will be used to categorize vital sign measurements observed during this clinical trial.

Observed values and changes from pre-injection (Baseline) to post-injection (at Day 1, 60 minutes after study intervention) for all vital sign measurements will be summarized by
vaccination group. A toxicity grade shift table of the vital signs from pre-injection to post-injection will be provided as well.

A listing containing individual participant vital sign measurement data will be provided. Additionally, participant with any abnormal post-baseline vital sign measurement where toxicity grade (Grade 3 or higher) will be listed separately: if a participant has a vital sign result with Grade 3 or higher abnormality after injection visit, then all results for that participant will be presented in the listing.

If multiple values are collected within a post-baseline visit/timepoint, the last assessment will be used in the by-visit summary tables. Unscheduled visits (including early termination) will not be summarized in by-visit summaries of data but may contribute to either baseline or post-baseline worst-case (maximum, minimum, etc.) values when applicable.

# 2.6.3.6. Pregnancy Testing

For participants of childbearing potential, a point-of-care urine pregnancy test will be performed at the Screening Visit and before injection at Day 1. At the discretion of the Investigator, a pregnancy test either via blood or point-of-care urine can be performed at any time. For participants of nonchildbearing potential, the FSH level may be measured at the Screening Visit, as necessary, and at the discretion of the Investigator, to confirm menopausal status.

A listing containing individual participant pregnancy test results will be provided for the pregnancy tests and FSH blood levels.

#### 2.6.3.7. Other Safety Data

# 2.6.3.7.1 Safety Telephone Calls

A safety telephone call is a telephone call made to the participant by trained site personnel. This call will follow a script, which will facilitate the collection of relevant safety information.

A listing containing individual participant safety call information will be provided.

# 2.6.3.7.2 Assessment for Respiratory Viral Infection

For Part 1, during the clinical trial, participants might experience symptoms consistent with ILI or SARS-CoV-2 infection. All participants will provide nasal swab samples before the injection on Day 1 for assessment of infection with respiratory pathogens, including influenza viruses and SARS-CoV-2, as influenza or COVID-19 symptoms may confound reactogenicity assessments. Throughout the clinical trial, the participant will be instructed to contact the study site if they have symptoms suggestive of ILI or SARS-CoV-2. An unscheduled visit for symptom assessment and nasal swab for viral respiratory pathogens will be conducted within 7 days of the onset of any potential ILI or SARS-CoV-2 symptoms.

The Assessment for Respiratory Viral Infection is available in protocol Section 8.3.7 corresponding to the Efficacy Analysis. A listing presenting for each participants the symptoms of ILI/COVID-19 will be provided as well.

# 2.6.3.7.3 Physical examination

A complete physical examination will include, at a minimum, assessments of skin, head, ears, eyes, nose, throat, neck, thyroid, lungs, heart, cardiovascular system, abdomen, lymph nodes, and musculoskeletal system and extremities. Height and weight will also be measured and recorded.

# 2.6.3.7.4 Electrocardiograms

For participants aged ≥18 to <51 only, a 12-lead ECG will be obtained at Day 1, after 10 minutes of supine rest. The purpose of the ECG is to serve as a Baseline comparison, should it be necessary, for subsequent clinical evaluation of suspected myocarditis and/or pericarditis. Clinically significant abnormal ECG findings, if incidentally observed by the Investigator, may contribute to Investigator's assessment of eligibility, at his or her discretion.

# 2.6.4. Immunogenicity Analysis

The primary analysis population for immunogenicity will be the PP Set. Planned timepoints for all immunogenicity assessments are provided in the SoA available in Appendix A.

For Part 1, the following analytes will be measured:

- Influenza: Serum antibody level as measured by HAI assay and potentially serum neutralizing antibody (nAb) level as measured by microneutralization assay.
- SARS-CoV-2: Serum nAb titers as measured by pseudovirus neutralization assay (PsVNA) assay and potentially serum binding antibody titers by enzyme-linked immunosorbent assay or multiplex assay specific to the SARS-CoV-2 proteins.
- Cellular immunogenicity in a subset of participants.

For secondary and exploratory endpoints, the Geometric Mean Titer (GMT) will be calculated using the following formula (Nauta, 2011):

$$2^{\left\{\frac{\sum_{i=1}^{n} log_2(t_i)}{n}\right\}}$$

where  $t_1, t_2, ..., t_n$  are *n* observed immunogenicity titers or levels.

The Geometric Mean Fold Rise (GMFR) measures the changes in immunogenicity titers or levels within participants. The GMFR will be calculated using the following formula:

$$2^{\left\{\frac{\sum_{i=1}^{n} log_{2}\binom{v_{ij}}{v_{ik}}}{n}\right\}} = 2^{\left\{\frac{\sum_{i=1}^{n} log_{2}(v_{ij}) - log_{2}(v_{ik})}{n}\right\}}$$

where, for *n* participants,  $v_{ij}$  and  $v_{ik}$  are observed immunogenicity titers or levels for participant *i* at time points *j* and *k*,  $j \neq k$ . For GMFR calculation, antibody values reported as below LLOQ will be replaced by LLOQ.

The 95% CIs for GMT and GMFR will be calculated based on the t distribution of the log-transformed values then back transformed to the original scale for presentation, unless otherwise specified.

### 2.6.4.1. Secondary Immunogenicity Endpoints

- GMT and GMFR at Day 29 compared with Day 1 by HAI assay for influenza and PsVNA for SARS-CoV-2
- Influenza: Percentage of participants with seroconversion, defined as a Day 29 titer CCI if Baseline is CCI or a 4-fold or greater rise if Baseline is CCI in anti-HA antibodies measured by HAI assay

- SARS-CoV-2: Percentage of participants with seroresponse, defined as a Day 29 titer
   ≥ 4-fold if Baseline is ≥ LLOQ or ≥ 4 × LLOQ if Baseline titer is < LLOQ in nAb</li>
   titers measured by PsVNA (or binding antibody assay)
- GMT and GMFR compared with Day 1 (Baseline) by HAI for influenza and PsVNA (or binding antibody assay) for SARS-CoV-2 at all evaluable timepoints
- Percentages of participants with seroconversion (influenza) and seroresponse (SARS-CoV-2) as defined below, at all evaluable timepoints

For the secondary immunogenicity endpoints, descriptive summaries statistics, including median, Q1, Q3, minimum, and maximum along with the number and percentage values above (>=) LLOQ and below (<) LLOQ will be provided for the antibody titer values by treatment arm (available in Section 2.6.1) for the influenza and SARS-CoV-2 endpoints. In addition, the following endpoints summaries will be provided:

- Geometric mean of specific antibody titers (GMT) with corresponding 2-sided 95%
   CI at each time point
- Geometric mean fold rise (GMFR) of specific antibody titers with the corresponding 2-sided 95% CI at each post-Baseline time point over pre-injection Baseline at Day 1,

Listing presenting the antibody level, for each specific strain of influenza and SARS-CoV-2 will be provided. The ratio of post-Baseline/Baseline, LLOQ and ULOQ will be presented as well. An additional listing will be provided for participants with Influenza or SARS-CoV-2 infections.

Reverse Cumulative Distribution Function for each specific strain of influenza and SARS-CoV-2 will be provided. The box plot for GMT and GMFR will be provided at all evaluable timepoints. The bar plot for GMFR at Day 29 will also be provided.

$$2^{\left\{\frac{\sum_{i=1}^{n} log_{2}(t_{i})}{n}\right\}} 2^{\left\{\frac{\sum_{i=1}^{n} log_{2}\binom{v_{ij}}{v_{ik}}}{n}\right\}} = 2^{\left\{\frac{\sum_{i=1}^{n} log_{2}(v_{ij}) - log_{2}(v_{ik})}{n}\right\}}$$

Additional descriptions will be provided by treatment arm (available in Section 2.6.1) for the following influenza and SARS-CoV-2 endpoints:

Percentages of participants with seroconversion (influenza) and seroresponse (SARS-CoV-2) with the corresponding 2-sided 95% CI at each post-Baseline time point,

• Percentages of participants with a GMFR results >=2, and >=4 with the corresponding 2-sided 95% CI at each post-Baseline time point.

For participants in the groups receiving mRNA-1083, mRNA-1010 or influenza injections, seroconversion rate from Baseline will be provided with a 2-sided 95% CI using the Clopper-Pearson method at each post-Baseline time point. Rate of seroconversion is defined as the proportion of participants with either a pre-vaccination HAI titer CCI and a post-vaccination HAI titer CCI or a pre-vaccination HAI titer CCI and a minimum 4-fold rise in post-vaccination HAI antibody titer.

For participants in the groups receiving mRNA-1083, mRNA-1283.222 or mRNA-1273.222, seroresponse rate will be summarized for planned post-Baseline visits, including the 2-sided 95% CI using the Clopper-Pearson method. Rate of Seroreponse for SARS-Cov-2 is defined as  $a \ge 4$  fold rise in nAb titer from Baseline in those with Baseline titer  $\ge$  LLOQ, or a post-Baseline titer  $\ge$  4 × LLOQ if Baseline titer is < LLOQ.

In addition, the following analysis statistics will be provided by treatment arm (available in Table 7) at Day 29 and D181 for the following influenza and SARS-CoV-2 endpoints:

- Within Treatment Group, Model-based geometric mean titer (GMT) with the corresponding 95% CI,
- Between Treatment Group, Pair-wise geometric mean ratios (GMR) with the corresponding 95% CI

The model-based GM titer will be estimated based on an analysis of covariance (ANCOVA) model, and it will be modelled separately for Cohort A and Cohort B. In the ANCOVA model, the log-transformed antibody titer at a post-Baseline timepoint (Day 29 or Day 181) are treated as a dependent variable, with the treatment group as an explanatory variable and covariates listed in Table 6 below for different assays, Cohorts and subgroups:

**Table 6 Covariates Included in Different ANCOVA Models (Part 1)** 

| Assay | Cohort | Subgroup | Covariate(s) |
|---|---|---|---|
| | | Overall | Influenza vaccine status since Sept 2022 (IRT) |
| | | Overall | None |
| | A | Prior bivalent Covid vaccine status: Received | None |
| | A | Prior bivalent Covid vaccine status: Not Received | None |
| | | Baseline SARS-CoV2 Status: Positive | None |
| | | Baseline SARS-CoV2 Status: Negative | None |
| PsVNA | | Overall | Age Group (IRT), Influenza vaccine status since Sept 2022 (IRT) |
| ISVINA | | Overall | Age Group (EDC) |
| | | Age Group (EDC): $\geq 18$ to $\leq 50$ years | None |
| | В | Age Group (EDC): $\geq 50$ to $<65$ years | None |
| | | Prior bivalent Covid vaccine status: Received | Age Group (IRT) |
| | | Prior bivalent Covid vaccine status: Not Received | Age Group (IRT) |
| | | Baseline SARS-CoV2 Status: Positive | Age Group (IRT) |
| | | Baseline SARS-CoV2 Status: Negative | Age Group (IRT) |
| | | Overall | Influenza vaccine status since Sept 2022 (IRT) |
| | A | Overall | Influenza vaccine status since Sept 2022 (EDC) |
| | A | Influenza vaccine status since Sept 2022 (EDC): Received | None |
| | | Influenza vaccine status since Sept 2022 (EDC): Not Received | None |
| HAI | | Overall | Age Group (IRT), Influenza vaccine status since Sept 2022 (IRT) |
| 117.11 | | Overall | Age Group (EDC), Influenza vaccine status since Sept 2022 (EDC) |
| | В | Age Group (EDC): $\geq 18$ to $<50$ years | Influenza vaccine status since Sept 2022 (IRT) |
| | | Age Group (EDC): $\geq$ 50 to <65 years | Influenza vaccine status since Sept 2022 (IRT) |
| | | Influenza vaccine status since Sept 2022 (EDC)=Y | Age Group (IRT) |
| | | Influenza vaccine status since Sept 2022 (EDC)=N | Age Group (IRT) |

The GMT will be estimated by the geometric least square mean (GLSM) from the ANCOVA model for each treatment group and corresponding 2-sided 95% CI will be provided.

For each pair of between-group comparison specified in Table 7, the GMR (ratio of GMTs) between the two treatment groups in each pair will be estimated from the ANCOVA model, with 2-sided 95% CI provided accordingly.

Additional comparisons or analysis statistics will be provided by treatment arm (available in Table 7) at Day 29 for the following influenza and SARS-CoV-2 endpoints:

• Pair-wise seroconversion rate (SCR) difference (influenza) and pair-wise seroresponse rate (SRR) difference (SARS-CoV-2) with the corresponding 95% CI

For each pair of between-group comparison specified in Table 7, the difference of seroresponse/seroconversion rate (SRR/SCR) between the two treatment groups in each pair at Day 29 will be provided, with 2-sided 95% CI estimated using Miettinen-Nurminen method.

A bar plot for GMR and GMFR at Day 29 and at D181, as well as a bar plot of SCR (influenza)/SRR (SARS-CoV-2) at Day 29 and D181 will be provided.

Table 7 Exploratory between-group Immunogenicity comparisons (Part 1)

| | Influenza Cohort A | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | Treatm | ent Arm | | | |
| Control<br>Arm | mRNA-<br>1010<br>μg | mRNA-<br>1010 μg | mRNA-<br>1083.1 μg | mRNA-<br>1083.1 μg | mRNA-<br>1083.2<br>μg | mRNA-<br>1083.2<br>μg | mRNA-<br>1083.2 μg | mRNA-<br>1083.3<br>CCI μg |
| Fluarix | X | X | X | X | X | X | X | X |
| Fluzone<br>HD | X | X | X | X | X | X | X | X |
| mRNA-<br>1010 μg | NA | X | X | X | X | X | X | X |
| mRNA-<br>1010. μg | NA | NA | X | X | X | X | X | X |

| | Influenza Cohort B | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | Tr | eatment A | rm | | | |
| Control<br>Arm | mRNA-<br>1010<br>μg | mRNA-<br>1010.<br>μg | mRNA-<br>1083.1<br>μg | mRNA-<br>1083.1<br>μg | mRNA-<br>1083.1<br>μg | mRNA-<br>1083.2<br>CCl μg | mRNA-<br>1083.2<br>μg | mRNA-<br>1083.2<br>μg | mRNA-<br>1083.3<br>CCI μg |
| Fluarix | X | X | X | X | X | X | X | X | X |
| mRNA-<br>1010 | | | | | | | | | |
| μg | NA | X | X | X | X | X | X | X | X |
| mRNA-<br>1010. μg | NA | NA | X | X | X | X | X | X | X |

| | SARS-CoV-2 Cohort A | | | | | | |
|---|---|---|---|---|---|---|---|
| | | Treatment Arm | | | | | |
| Control Arm | mRNA-<br>1283.222<br>μg | mRNA-<br>1083.1<br>μg | mRNA-<br>1083.1<br>μg | mRNA-<br>1083.2<br>CCI μg | mRNA-<br>1083.2<br>μg | mRNA-<br>1083.2<br>μg | mRNA-<br>1083.3<br>CCI μg |
| mRNA-<br>1273.222 μg | X | X | X | X | X | X | X |
| mRNA-<br>1283.222 μg | NA | X | X | X | X | X | X |

| | SARS-CoV-2 Cohort B | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Treatment Arm | | | | | | |
| | mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- mRNA- <th< th=""><th>mRNA-<br/>1083.3</th></th<> | | | | | | | mRNA-<br>1083.3 |
| Control Arm | μg | <mark>ccι</mark> μg | <mark>ccl</mark> μg | <mark>ccl</mark> μg | <mark>CCI</mark> μg | <mark>ccl</mark> μg | <mark>ccl</mark> μg | <mark>CCI</mark> μg |
| mRNA-<br>1273.222 μg | X | X | X | X | X | X | X | X |
| mRNA-<br>1283.222 μg | NA | X | X | X | X | X | X | X |

# 2.6.4.2. Exploratory Immunogenicity Endpoints

The below exploratory analyses of immunogenicity may be performed:

• GMT and GMFR (compared to Day 1) to vaccine mismatched strains at all evaluable time points

- GMT and GMFR (compared to Day 1) to vaccine matched and mismatched strains assayed by alternative methods (including but not limited to: microneutralization assay for influenza or ligand-binding assay for SARS-CoV-2) at all evaluable time points
- Frequency, magnitude, and phenotype of virus specific T-cell and B-cell responses measured by flow cytometry or other methods, and to perform targeted repertoire analysis of B cells and T cells after vaccination
- Frequency, specificities, or other endpoints to be determined for the further characterization of immune responses

### 2.6.5. Exploratory Analysis

# 2.6.5.1. Efficacy Analysis

While the study will not be powered for efficacy assessments, symptoms of infection with respiratory pathogens will be tracked as an exploratory objective in this study (Part 1 only). Efficacy analyses will be performed on the FAS. Frequency of RT-PCR-confirmed protocoldefined influenza-like illness (ILI) and RT-PCR-confirmed symptomatic SARS-CoV-2 observed among the participants in the FAS will be summarized according to the vaccination groups as randomized.

### 2.6.5.2. Influenza Infection

A protocol-defined ILI is determined by the occurrence of at least 1 respiratory illness symptom concurrently with at least 1 systemic symptom, or the occurrence of any 2 or more respiratory symptoms, as shown in Table 8.

An RT-PCR confirmed protocol-defined ILI is defined as a positive influenza result on a respiratory sample by RT-PCR performed at the Global Central Laboratory and/or a local certified laboratory within 7 days of onset of protocol-defined ILI at any time during the study period.

Table 8 Respiratory and Systemic Symptoms for Protocol-defined ILI (Part 1)

| Respiratory symptoms | Systemic symptoms |
|---|---|
| Sore throat | Body temperature ≥37.5°C [≥99.5°F] |
| Cough/rhinorrhea/nasal congestion (≥1 of | Chills |
| the 3 symptoms count as 1 respiratory | Tiredness |
| symptom) | Headache |
| Sputum production | Myalgia |
| Wheezing | Nausea/vomiting |
| Difficulty breathing | Diarrhea |

Derivation of PT-PCR confirmed protocol-defined ILI:

The eligible protocol-defined ILI symptoms will be documented on the ILI symptom assessment eCRF. The following derivation steps will be performed on each participant to determine whether protocol-defined ILI occurred within the specified window based on positive RT-PCR results:

Step 1: The time window for protocol-defined ILI to be considered as RT-PCR confirmed will be calculated based on each positive RT-PCR collection date +/- 7 days (ex: positive RT-PCR collection date - 7 days through positive RT-PCR collection date + 7 days).

Step 2: Within this time window, determine the earliest eligible symptoms for protocol-defined ILI. Considering the symptoms listed in (Table 8) that onset within the positive RT-PCR collection date window from Step 1, eligible symptoms are defined as those that meet either of the criteria given below, based on their start and end dates:

- The occurrence of at least 1 respiratory illness symptom and at least 1 systemic symptom that overlap for at least 1 day or
- The occurrence of any 2 or more respiratory symptoms that overlap for at least 1 day.

Step 3: The start date for the RT-PCR confirmed protocol-defined ILI will be set as either the positive RT-PCR date or the earliest eligible symptom onset date, whichever occurs earlier.

The following summaries will be provided for influenza infection:

• The number and percentage of participants with an RT-PCR test results (Positive, Negative, Not Applicable, Missing) at Baseline will be summarized by vaccination group (as defined in Section 2.6.1).


- The number and percentage of participants with an RT-PCR test results (Positive, Positive and <=14 Days After Injection, Positive and > 14 Days After Injection, Negative, Not Applicable, Missing) excluding Baseline will be summarized by vaccination group (as defined in Section 2.6.1).
- The number and percentage of participants with RT-PCR confirmed protocol-defined ILI within the period starting from 14 days post-injection up through EoS will be summarized by strain of influenza virus, and by time period. A 2-sided 95% CI using the Clopper-Pearson method will be provided for the percentage of participants with the RT-PCR confirmed influenza infection.
- The number and percentage of participants with RT-PCR confirmed protocol-defined ILI within the period starting from 14 days post-injection up through EoS will be summarized by respiratory symptoms and systemic symptoms
- A listing presenting the RT-PCR test results for influenza will be provided.
- A listing presenting the symptom assessment for protocol-defined ILI will be provided.

#### 2.6.5.3. SARS-CoV-2 Infection

Symptomatic COVID-19 is defined by the presence of one of the CDC-listed symptoms (CDC, 2020) and a positive RT-PCR test on a respiratory sample. SARS-CoV-2 should be suspected if the participant experiences any one of the symptoms listed below lasting at least 48 hours (except for fever and/or respiratory symptoms) (CDC, 2020):

- Fever (temperature ≥38.0°C [100.4°F]) or chills (of any duration, including ≤48 hours)
- Cough (of any duration, including ≤48 hours)
- Shortness of breath and/or difficulty breathing (of any duration, including ≤48 hours)
- Fatigue
- Muscle or body aches
- Headache
- New loss of taste and/or smell
- Sore throat, congestion, or runny nose
- Nausea or vomiting

#### Diarrhea

Symptomatic COVID-19 is defined by the presence of one of the CDC-listed symptoms (CDC, 2020) and a positive RT-PCR test on a respiratory sample.

If the participant had known exposure to COVID-19 (eg, exposure to someone with a confirmed case of COVID-19), it will be captured in the COVID-19 exposure form, and the participant will continue to follow all remaining study assessments as scheduled. Likewise, participants with a confirmed case of COVID-19 will continue to follow all remaining study assessments as scheduled.

The following summaries will be provided:

- The number and percentage of participants with an RT-PCR test results (Positive, Negative, Not Applicable, Missing) at Baseline will be summarized by vaccination group (as defined in Section 2.6.1).
- The number and percentage of participants with an RT-PCR test results (Positive, Positive and <=14 Days After Injection, Positive and > 14 Days After Injection, Negative, Not Applicable, Missing) excluding Baseline will be summarized by vaccination group (as defined in Section 2.6.1).
- The number and percentage of participants with, and the number of events of RT-PCR confirmed SARS-CoV-2 Infection, and RT-PCR Symptomatic SARS-CoV-2 Infection within the period starting from 14 days post-injection up through EoS will be summarized by time period.
- A listing presenting the RT-PCR test results for SARS-CoV-2 infection will be provided.
- A listing presenting the symptom assessment for SARS-CoV-2 infection will be provided.

# 2.6.6. Other Exploratory Endpoints

Transcriptomic and genomic samples will be part of the optional biomarker assessment. Exploratory assessments may include assessment of biomarkers for safety, reactogenicity, and inflammation. Serologic markers of disease severity, immune response to SARS-CoV-2 or influenza, RT-PCR of nasal swab samples, genetic sequences of SARS-CoV-2 or influenza

strains isolated from participants' samples, and genomic and transcriptomic samples may also be evaluated. Analyses and reporting of these endpoints will be covered in a separate analysis plan if applicable.

# 2.6.7. Planned Analyses

# 2.6.7.1. Interim Analysis

An interim analysis of safety, reactogenicity, and immunogenicity is planned after all the participants in Cohort A and B have completed the Day 29 visit. The interim analysis as of completion of Day 29 will be performed by the study statistician and programmers. The group-level unblinded summary data of the Day 29 interim analyses may be reviewed by the Sponsor project team for safety monitoring and/or clinical development planning purposes for the mRNA-1083 project. More details will be documented in the study Data Blinding Plan.

In addition, another interim analysis for reactogenicity data up to Day 8 only may be performed after all the participants in Cohort A and B have completed the Day 8 visit. The potential interim analysis as of completion of Day 8 may be performed by an independent team of unblinded statistician and programmers. More details will be documented in the study Data Blinding Plan.

### 2.6.7.2. Final Analysis

The final analysis will be performed after all the participants in both Cohort A and Cohort B have completed the Day 181/EoS visit.

#### 3. Part 2

# 3.1. Study Objectives

# 3.1.1. Primary Objectives

The primary objectives are:

- To evaluate the safety and reactogenicity of study intervention administration across study treatment arms
- To evaluate the humoral immune responses to vaccine-matched strains for influenza and SARS-CoV-2 across study treatment arms at Day 29

# 3.1.2. Secondary Objectives

The secondary objective is:

 To evaluate the humoral immune responses to vaccine-matched strains for influenza and SARS-CoV-2 across study treatment arms at all evaluable humoral immunogenicity time points

# 3.1.3. Exploratory Objectives

The following exploratory objectives may be assessed:

- To evaluate the humoral immune responses to vaccine-mismatched strains for influenza and SARS-CoV-2 across study treatment arms
- To evaluate the humoral immune responses against vaccine-matched and vaccine-mismatched strains for influenza and SARS-CoV-2 across study treatment arms
- To further characterize the immune response to influenza and SARS-CoV-2 across study treatment arms

# 3.2. Study Endpoints

# 3.2.1. Primary Endpoints

• Solicited local and systemic ARs through 7 days after injection

- Unsolicited AEs through 28 days after injection
- Unsolicited Severe AEs through 28 days after injection
- Unsolicited MAAEs from Day 1 to Day 181/EoS
- Unsolicited AESIs from Day 1 to Day 181/EoS
- SAEs from Day 1 to Day 181/EoS
- Unsolicited AEs leading to discontinuation from Day 1 to Day 181/EoS
- GMT and GMFR at Day 29 compared to Day 1 by HAI assay for influenza and by PsVNA for SARS-CoV-2
- Influenza: Percentage of participants with seroconversion, defined as a Day 29 titer CCI if Baseline is CCI or a 4-fold or greater rise if Baseline is CCI in anti-HA antibodies measured by HAI assay
- SARS-CoV-2: Percentage of participants with seroresponse, defined as a Day 29 titer
   ≥4-fold if Baseline is ≥LLOQ or ≥4 × LLOQ if Baseline titer is <LLOQ in nAb titers</li>
   measured by PsVNA

# 3.2.2. Secondary Endpoints

- GMT and GMFR at all evaluable time points compared to Day 1 by HAI for influenza and PsVNA for SARS-CoV-2
- Influenza: Percentage of participants with seroconversion, as defined in Section 3.2.1
- SARS-CoV-2: Percentage of participants with seroresponse, as defined in Section 3.2.1

#### 3.2.3. Exploratory Endpoints

- GMT and GMFR at all evaluable time points compared to Day 1 by HAI for influenza and PsVNA for SARS-CoV-2
- Influenza: Percentage of participants with seroconversion, as defined in Section 3.2.1
- SARS-CoV-2: Percentage of participants with seroresponse, as defined in Section 3.2.1

- GMT and GMFR at all evaluable time points compared to Day 1 by alternative methods, including, but not limited to: microneutralization assay for influenza or ligand-binding assay for SARS-CoV-2
- Frequency, specificities, or other endpoints to be determined for the further characterization of immune responses

# 3.3. Study Design

# 3.3.1. Overall Study Design

Part 2 of the study will be a Phase 2 randomized, stratified, observer-blind, active-control study to evaluate the safety, reactogenicity, and immunogenicity of mRNA-1083 compositions and dose levels compared with active-control vaccines mRNA-1010, mRNA-1283.815, mRNA-1273.815, and licensed active-control vaccine, Fluarix in healthy adults ≥18 to <50 years of age. Approximately 520 participants ≥18 to <50 years of age will be enrolled. Participants will be randomized (in equal allocation ratio) into the investigational treatment arms, stratified by influenza vaccine status in the most recent influenza season (received or not received since Sept 2023). Table 9 lists the details of study cohorts and dose levels for study vaccine administration. All participants will receive a single IM injection of study intervention administered in a deltoid muscle on Day 1.

Table 9 Study Arm(s) and Interventions (Part 2)

| Part 2 Arm:<br>(≥18 to <50 years),<br>n=40/arm, 520 total | Intervention | Total mRNA<br>Dose (μg) <sup>a</sup> | Intervention<br>Type |
|---|---|---|---|
| 1 | mRNA-1083 CCI | CCI | IP |
| 2 | mRNA-1083 | | IP |
| 3 | mRNA-1083 | | IP |
| 4 | mRNA-1083 | | IP |
| 5 | mRNA-1083 | | IP |
| 6 | mRNA-1083 | | IP |
| 7 | mRNA-1083 | | IP |
| 8 | mRNA-1083 | | IP |
| 9 | mRNA-1010 CC | | Non-IP experimental comparator |
| 10 | mRNA-1010 | | Non-IP experimental comparator |
| 11 | mRNA-1283.815 | | Non-IP experimental comparator |
| 12 | mRNA-1273.815 | | Licensed vaccine comparator |
| 13 | Fluarix | - | Licensed vaccine comparator |

All participants of the study will participate in a Screening period (up to 28 days before Day 1), treatment period (single dose of vaccine on Day 1), and a follow-up period (up to 6 months after vaccination). The study schema is presented in Figure 2 Study Schema. Please refer to the Part 2 Schedule of Activities (SoA) available in Appendix A.

Figure 2 Study Schema (Part 2)



Abbreviation: mRNA = messenger ribonucleic acid

# 3.3.2. Statistical Hypotheses

See Section 2.3.2 for details.

# 3.3.3. Sample Size and Power

Approximately, 520 participants will be enrolled at an evenly allocated ratio across the 13 treatment arms for adults  $\geq$ 18 to <50 years of age, with 40 participants planned for each arm. Approximately 40 participants in each group receiving an investigational injection have approximately 80.5% (or 87.1%) probability to observe at least 1 participant with an AE given the true underlying incidence rate of AE is 4% (or 5%) (Table 10).


**Table 10 Sample Size Determination (Part 2)** 

| Sample Size | True AE Rate | Probability of 0 AEs | Power to Detect at Least 1 AE |
|---|---|---|---|
| 40 | 2.0% | 44.6% | 55.4% |
| 40 | 3.0% | 29.6% | 70.4% |
| 40 | 4.0% | 19.5% | 80.5% |
| 40 | 5.0% | 12.9% | 87.1% |

#### 3.3.4. Randomization

Participants will be randomized (in equal allocation ratio) into the investigational treatment arms, stratified by influenza vaccine status in the most recent influenza season (received or not received since Sept 2023).

# 3.4. Blinding and Unblinding

The planned analyses including a Day 29 interim analysis are described in Section 3.6.6 of this SAP. For further details on preidentified sponsor and CRO team members (identified by role), and the level of unblinding (treatment group level unblinding and/or subject level unblinding) at the IAs and the Final analysis, please refer to the study Data Blinding Plan.

#### 3.5. Analysis Sets

#### 3.5.1. Randomization Set

See Section 2.5.1 for details.

# 3.5.2. Full Analysis Set (FAS)

See Section 2.5.2 for details.

#### 3.5.3. Per Protocol (PP) Set

The PP Set in Part 2 consists of all participants in the FAS who comply with the injection schedule, comply with the timings of immunogenicity blood sampling to have a Baseline and at least 1 post-injection assessment at Day 29 (-7 to +14 days), have no documented infection (confirmed by RT-PCR test) of either influenza or SARS-CoV-2 on Day 1, have no major dosing error, and have no major protocol deviations or conditions/medications that affect the immune

response. The PP Set will be used as the primary analysis set for analyses of immunogenicity unless otherwise specified. Participants will be analyzed according to the group to which they were randomized.

The major dosing error ranges, available in Table 11, will be used to determine participant exclusion from the PP analysis populations:

**Table 11 Exclusion Condition for Dosing Errors (Part 2)** 

| Randomized Group | <b>Exclusion Conditions</b> |
|---|---|
| mRNA-1083 CCI ( <sup>CCI</sup> μg) | Any of the following received: mRNA-1083 CCI ≤ CCI μg OR mRNA-1083 CCI > CCI μg OR mRNA-1083 OR mRNA-1010 OR mRNA-1283.815 OR mRNA-1273.815 OR Fluarix |
| mRNA-1083 CCI ( <sup>CCI</sup> μg) | Any of the following received: mRNA-1083 CCI ≤ COI μg OR mRNA-1083 CCI > COI μg OR mRNA-1083 OR mRNA-1010 OR mRNA-1283.815 OR mRNA-1273.815 OR Fluarix |
| mRNA-1083 CCI ( <sup>CCI</sup> μg) | Any of the following received: mRNA-1083 CCI ≤ μg OR mRNA-1083 CCI > CCI μg OR mRNA-1083 OR mRNA-1010 OR mRNA-1283.815 OR mRNA-1273.815 OR Fluarix |
| mRNA-1083 CCI ( μg) | Any of the following received: mRNA-1083 CCI ≤ μg OR mRNA-1083 CCI > μg OR mRNA-1083 OR mRNA-1010 OR mRNA-1283.815 OR mRNA-1273.815 OR Fluarix |
| mRNA-1083 CCI ( <sup>CCI</sup> μg) | Any of the following received: mRNA-1083 CCI ≤ COI μg OR mRNA-1083 CCI > COI μg OR mRNA-1083 OR mRNA-1010 OR mRNA-1283.815 OR mRNA-1273.815 OR Fluarix |
| mRNA-1083 CCI ( μg) | Any of the following received: mRNA-1083 CCI ≤ COI μg OR mRNA-1083 CCI > COI μg OR mRNA-1083 OR mRNA-1010 OR mRNA-1283.815 OR mRNA-1273.815 OR Fluarix |
| mRNA-1083 CCI ( <sup>CCI</sup> μg) | Any of the following received: mRNA-1083 CCI ≤ μg OR mRNA-1083 CCI > CCI μg OR mRNA-1083 OR mRNA-1010. OR mRNA-1283.815 OR mRNA-1273.815 OR Fluarix |
| mRNA-1083 CCI ( μg) | Any of the following received: mRNA-1083 CCI ≤ μg OR mRNA-1083 CCI > μg OR mRNA-1083 OR mRNA-1010 OR mRNA-1283.815 OR mRNA-1273.815 OR Fluarix |
| mRNA-1010. ( <sup>CCI</sup> μg) | Any of the following received: mRNA-1010 μg OR mRNA-1010 γ μg OR mRNA-1083 CC OR mRNA-1083 CC OR mRNA-1283.815 OR mRNA-1273.815 OR Fluarix |
| mRNA-1010. ( <sup>CC</sup> μg) | Any of the following received: mRNA-1010 |
| mRNA-1283.815 ( <sup>CCI</sup> μg) | Any of the following received:<br>mRNA-1283.815 ≤ μg OR mRNA-1283.815 > μg OR |

| Randomized Group | Exclusion Conditions |
|---|---|
| | mRNA-1083 CCI OR mRNA-1083 CCI OR mRNA-1010. OR mRNA-1273.815 OR Fluarix |
| DNIA 1272 915 (CO) | |
| mRNA-1273.815 ( μg) | Any of the following received: |
| | mRNA-1273.815 ≤ μg OR mRNA-1273.815 > μg OR mRNA-1083 CCI OR mRNA-1010. OR |
| | mRNA-1083 CCI OR mRNA-1083 CCI OR mRNA-1010. OR |
| | mRNA-1283.815 OR Fluarix |
| Fluarix | Any of the following received: |
| | Fluarix ≤ 30 μg OR |
| | mRNA-1083 CCI OR mRNA-1083 CCI OR mRNA-1010 OR mRNA- |
| | 1283.815 OR mRNA-1273.815 |

# 3.5.4. Safety Set

See Section 2.5.4 for details. Participants will be included in the vaccination group corresponding to what they actually received according to the as treated scheme given below in Table 12.

**Table 12 As Treated Grouping Scheme (Part 2)** 

| Group Name | Inclusion condition |
|---|---|
| mRNA-1083 CCI ( <sup>cci</sup> μg) | Any dose of mRNA-1083 CC > CC μg |
| mRNA-1083 ( <sup>CCI</sup> μg) | Any dose of mRNA-1083 $>$ CCI $\mu g$ and $\leq$ CCI $\mu g$ |
| mRNA-1083 ( <sup>CCI</sup> μg) | Any dose of mRNA-1083 $\rightarrow$ $\mu g$ and $\leq$ $\mu g$ |
| mRNA-1083 (μg) | Any dose of mRNA-1083 ≤ μg |
| mRNA-1083 ( <sup>cct</sup> μg) | Any dose of mRNA-1083 > CCI μg |
| mRNA-1083 ( <sup>CCI</sup> μg) | Any dose of mRNA-1083 $>$ CCI $\mu g$ and $\leq$ CCI $\mu g$ |
| mRNA-1083 ( <sup>CCI</sup> μg) | Any dose of mRNA-1083 $\rightarrow$ $\mu g$ and $\leq$ $\mu g$ |
| mRNA-1083 (μg) | Any dose of mRNA-1083 ≤ μg |
| mRNA-1010 $(\frac{\omega}{\mu}g)$ | Any dose of mRNA-1010 $\sim \frac{1}{\mu g}$ |
| mRNA-1010. (μg) | Any dose of mRNA-1010. ≤ □ μg |
| mRNA-1283.815 ( <sup>CCI</sup> μg) | Any dose of mRNA-1283.815 |
| mRNA-1273.815 ( <sup>CCI</sup> μg) | Any dose of mRNA-1273.815 |
| Fluarix | Any dose of Fluarix |

# 3.5.5. Solicited Safety Set

See Section 2.5.5 for details.

# 3.6. Statistical Analysis

The SoA is provided in the Appendix A.

# 3.6.1. General Considerations

See Section 2.6.1 for details.

For calculation regarding antibody levels/titers, antibody values reported as below the lower limit of quantification (LLOQ) will be replaced by 0.5 × LLOQ. Values reported as above the upper limit of quantification (ULOQ) will be converted to the ULOQ. Missing results will not be imputed.

**Table layouts** will be presented according to vaccination group. First for the overall participants, then by subgroups as given in Table 13.

For Part 2, the following vaccination groups will be used for summary purposes for tables and figures outputs:

- Fluarix
- mRNA-1010. μg
- mRNA-1010. μg
- mRNA-1273.815 <sup>CCI</sup> μg
- mRNA-1283.815 μg
- mRNA-1083 **CCI** μg
- mRNA-1083 CCI <sup>CCI</sup> μg
- mRNA-1083 CCI α μg
- mRNA-1083 CCI <sup>CCI</sup> μg
- mRNA-1083 CCI μg
- mRNA-1083 CCI <sup>cci</sup> μg
- mRNA-1083 CCI <sup>CCI</sup> μg
- mRNA-1083 CCI <sup>CCI</sup> μg
- All mRNA-1083 CCI (all mRNA-1083 CCI vaccination groups combined; applicable to safety and reactogenicity analyses only)
- All mRNA-1083 CCI (all mRNA-1083 CCI vaccination groups combined; applicable to safety and reactogenicity analyses only)
- Overall (All vaccination groups combined; details are available below)

The "Overall" combined group will be presented for baseline summaries such as participant disposition, demographic summaries, concordance of randomization stratum, etc. as well as

major protocol deviation, medical history, concomitant medication and study duration summaries.

**Subgroups**: For Part 2, the following subgroups will be used for summary purposes, where indicated in this SAP. Unless otherwise specified, all subgroups are based on eCRF.

**Table 13 Definition for Subgroups (Part 2)** 

| Subgroup Variable | Categories |
|------------------------------------------|--------------|
| Influenza Vaccine Status Since Sept 2023 | Received |
| _ | Not Received |
| Covid Vaccine Status Since Sept 2023 | Received |
| | Not Received |
| Baseline SARS-CoV-2 Status | Positive |
| | Negative |

# 3.6.2. Background Characteristics

# 3.6.2.1. Participant Disposition

See Section 2.6.2.1 for details.

# 3.6.2.2. Demographics and Baseline Characteristics

Descriptive statistics for age, weight, height, and BMI are described in Section 2.6.2.2.

The number and percentage of participants will be provided for the following categorical variables:

- Sex (Male, Female)
- Race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, Multiracial, Other, Not Reported, Unknown)
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino, Not Reported, Unknown)
- Influenza vaccine status in the most recent influenza season (received or not received since Sept 2023) per eCRF
- Covid vaccine status (received or not received since Sept 2023) per eCRF
- Childbearing Potential for female participants (Yes/No) and reason if "No"
- Baseline SARS-CoV-2 RT-PCR Results (positive, negative, or missing)
- Baseline Elecsys Anti-SARS-CoV2 Results (positive, negative, or missing)

• Baseline SARS-CoV-2 Status (positive, negative, or missing)

The summaries will be provided separately for all analysis sets (except Randomization Set and Solicited Safety Set) defined in the Section 3.5. The number and percentage of participants randomized by country and site will be provided as well.

# 3.6.2.3. Medical History

See Section 2.6.2.3 for details.

### 3.6.2.4. Prior and Concomitant Medications

See Section 2.6.2.4 for details.

# 3.6.2.5. Study Exposure

See Section 2.6.2.5 for details.

# 3.6.2.6. Major Protocol Deviations

See Section 2.6.2.6 for details.

#### 3.6.3. Safety Analysis

See Section 2.6.3 for details.

#### 3.6.3.1. Solicited Adverse Reactions

See Section 2.6.3.1 for details.

#### 3.6.3.1.1 Overview of Solicited ARs

See Section 2.6.3.1.1 for details.

# 3.6.3.1.2 Solicited ARs by Toxicity Grade

See Section 2.6.3.1.2 for details.

# 3.6.3.1.3 Solicited ARs by Onset Day

See Section 2.6.3.1.3 for details.

#### 3.6.3.1.4 Characteristics of Solicited ARs

See Section 2.6.3.1.4 for details.

#### 3.6.3.1.5 Other solicited ARs summaries

See Section 2.6.3.1.5 for details.

# 3.6.3.2. Unsolicited Treatment-Emergent Adverse Events

See Section 2.6.3.2 for details.

Unsolicited AEs will be coded according to Medical Dictionary for Regulatory Activities (MedDRA) version 26.0 or higher and presented by MedDRA system organ class (SOC) and preferred term (PT).

SOC will be displayed in an internationally agreed order. PT will be displayed in descending order of frequency of the combined mRNA-1083 (CCI).

# 3.6.3.2.1 Overview of Unsolicited TEAEs

See Section 2.6.3.2.1 for details.

# 3.6.3.2.2 TEAEs by System Organ Class and Preferred Term

See Section 2.6.3.2.2 for details.

# 3.6.3.2.3 TEAEs by Preferred Term

Tables of all unsolicited TEAEs will be provided by PT sorted in a descending order starting with the frequency of the combined mRNA-1083 (CCI).

# 3.6.3.2.4 TEAEs by Severity

See Section 2.6.3.2.4 for details.

# 3.6.3.3. Death

See Section 2.6.3.3 for details.

### **3.6.3.4. Vital Signs**

See Section 2.6.3.5 for details.

# 3.6.3.5. Pregnancy Testing

See Section 2.6.3.6 for details.

# 3.6.3.6. Other Safety Data

# 3.6.3.6.1 Safety Telephone Calls

See Section 2.6.3.7.1 for details.

# 3.6.3.6.2 Assessment for Respiratory Viral Infection

For Part 2, all participants will provide nasal swab samples before the injection on Day 1 for assessment of infection with respiratory pathogens, including influenza viruses and SARS-CoV-2, as influenza or COVID-19 symptoms may confound reactogenicity assessments.

#### 3.6.3.6.3 Physical examination

See Section 2.6.3.7.3 for details.

# 3.6.3.6.4 Electrocardiograms

See Section 2.6.3.7.4 for details.

# 3.6.4. Immunogenicity Analysis

The primary analysis population for immunogenicity will be the PP Set. Planned timepoints for all immunogenicity assessments are provided in the SoA available in Appendix A.

For Part 2, the following analytes will be measured:

• Influenza: Serum antibody level as measured by HAI assay and potentially serum neutralizing antibody (nAb) level as measured by microneutralization assay.

• SARS-CoV-2: Serum nAb titers as measured by pseudovirus neutralization assay (PsVNA) assay and potentially serum binding antibody titers by enzyme-linked immunosorbent assay or multiplex assay specific to the SARS-CoV-2 proteins.

See section 2.6.4 for primary, secondary and exploratory endpoints calculation methods.

# 3.6.4.1. Primary Immunogenicity Endpoints

- GMT and GMFR at Day 29 compared to Day 1 by HAI assay for influenza and by PsVNA for SARS-CoV-2
- Influenza: Percentage of participants with seroconversion, defined as a Day 29 titer if Baseline is CCI or a 4-fold or greater rise if Baseline is CCI in anti-HA antibodies measured by HAI assay
- SARS-CoV-2: Percentage of participants with seroresponse, defined as a Day 29 titer
   ≥ 4-fold if Baseline is ≥ LLOQ or ≥ 4 × LLOQ if Baseline titer is < LLOQ in nAb
   titers measured by PsVNA</li>

For the primary immunogenicity endpoints, descriptive summaries statistics, including median, Q1, Q3, minimum, and maximum will be provided at Day 29 for the antibody titer values by treatment arm (available in Section 3.6.1) for the influenza and SARS-CoV-2 endpoints:

- GMT with corresponding 2-sided 95% CI
- GMFR of specific antibody titers with the corresponding 2-sided 95% CI at Day 29 over pre-injection Baseline at Day 1,

In addition, the following analysis statistics will be provided by treatment arm at Day 29 for the influenza and SARS-CoV-2 endpoints:

- Within treatment group, model-based GMT with the corresponding 95% CI,
- Between treatment group, pair-wise geometric mean ratios (GMR) with the corresponding 95% CI

The model-based GMT will be estimated by the geometric least square mean (GLSM) from the ANCOVA model for each treatment group and corresponding 2-sided 95% CI will be provided. In the ANCOVA model, the log-transformed antibody titer at Day 29 is treated as a dependent variable, with the treatment group as an explanatory variable and covariates listed in Table 14 for different assays and subgroups.

**Table 14 Covariates Included in Different ANCOVA Models (Part 2)** 

| Assay | Subgroup | Covariate(s) |
|---|---|---|
| | Overall | Log-transformed baseline antibody value,<br>Influenza Vaccine Status Since Sept 2023<br>(IRT) |
| | Overall | Log-transformed baseline antibody value |
| PsVNA | Covid Vaccine Status Since Sept 2023: Received | Log-transformed baseline antibody value |
| | Covid Vaccine Status Since Sept 2023: Not Received | Log-transformed baseline antibody value |
| | Baseline SARS-CoV2 Status: Positive | Log-transformed baseline antibody value |
| | Baseline SARS-CoV2 Status: Negative | Log-transformed baseline antibody value |
| | Overall | Log-transformed baseline antibody value,<br>Influenza Vaccine Status Since Sept 2023<br>(IRT) |
| HAI | Overall | Log-transformed baseline antibody value,<br>Influenza Vaccine Status Since Sept 2023<br>(EDC) |
| | Influenza Vaccine Status Since Sept 2023 (EDC): Received | Log-transformed baseline antibody value |
| | Influenza Vaccine Status Since Sept 2023 (EDC):<br>Not Received | Log-transformed baseline antibody value |

For each pair of between-group comparison specified in Table 15, the GMR between the two treatment groups in each pair will be estimated from the ANCOVA model, with its 2-sided 95% CI provided accordingly.

Seroconversion rate (SCR) for influenza from Baseline will be summarized at Day 29 with its 2-sided 95% CI using the Clopper-Pearson method for participants in the groups receiving mRNA-1083, mRNA-1010 or Fluarix.

• SCR at Day 29 is defined as the percentage of participants with a Day 29 titer CCI if Baseline is CCI or a 4-fold or greater rise if Baseline is CCI in anti-HA antibodies measured by HAI assay

Seroresponse rate (SRR) for SARS-CoV-2 from Baseline will be summarized at Day 29 with its 2-sided 95% CI using the Clopper-Pearson method for participants in the groups receiving mRNA-1083, mRNA-1283.815 or mRNA-1273.815.

SRR at Day 29 is defined as the proportion of participants with a Day 29 titer ≥ 4-fold
if Baseline is ≥ LLOQ or ≥ 4 × LLOQ if Baseline titer is < LLOQ in nAb titers
measured by PsVNA.</li>

Additional comparisons or analysis statistics will be provided by treatment arm at Day 29 for the influenza and SARS-CoV-2 endpoints. For each pair of between-group comparison specified in Table 15, the difference of seroresponse/seroconversion rate (SRR/SCR) between the two treatment groups in each pair will be provided, with its 2-sided 95% CI estimated using Miettinen-Nurminen method.

SCR, SRR, GM levels, GMFR and GMR will be plotted at Day 29: Reverse Cumulative Distribution Function for each specific strain of influenza and SARS-CoV-2 will be provided, as well as box plot and bar plot for GMT and GMFR, and bar plot for GMR, SCR and SRR.

Listing presenting the antibody level, for each specific strain of influenza and SARS-CoV-2 will be provided. The ratio of post-Baseline/Baseline, LLOQ and ULOQ will be presented as well.


Table 15 Between-group Immunogenicity comparisons (Part 2)

| | | | | Influenza | Compariso | ons | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Treatment Arm | | | | | | | | | |
| | | mRNA-<br>1010 μg | mRNA-<br>1010 μg | mRNA-<br>1083<br>(ΣΕ)<br>μg | mRNA-<br>1083<br>(ΣΕ)<br>μg | mRNA-<br>1083<br>(ΣΕ)<br>μg | mRNA-<br>1083<br>(CCI)<br>μg | mRNA-<br>1083<br>(CC)<br>μg | mRNA-<br>1083<br>(CC)<br>μg | mRNA-<br>1083<br>(CCI)<br>μg | mRNA-<br>1083<br>(CCI)<br>μg |
| Control Group | Fluarix | X | X | X | X | X | X | X | X | X | X |
| | mRNA-1010. μg | NA | X | X | X | X | X | X | X | X | X |
| | mRNA-1010. | NA | NA | X | X | X | X | X | X | X | X |
| | <u> </u> | | | SARS-CoV | -2 Compari | sons | | | • | | |
| | | | | Treatment Arm | | | | | | | |
| | | mRNA-1283.815 μg | | mRNA-<br>1083<br>(CC)<br>μg | mRNA-<br>1083<br>( μg | mRNA-<br>1083<br>( <sup>CCI</sup> )<br>μg | mRNA<br>-1083<br>(CCI)<br>μg | mRNA-<br>1083<br>(CC)<br>μg | mRNA-<br>1083<br>(CC)<br>μg | mRNA-<br>1083<br>(CCI)<br>μg | mRNA-<br>1083<br>(CCI)<br>μg |
| Group | mRNA-1273.815<br>μg | X | | X | X | X | X | X | X | X | X |
| Control Group | mRNA-1283.815<br>μg | NA | | X | X | X | X | X | X | X | X |

# 3.6.4.2. Secondary Immunogenicity Endpoints

- GMT and GMFR at all evaluable time points compared to Day 1 by HAI for influenza and PsVNA for SARS-CoV-2
- Influenza: Percentage of participants with seroconversion
- SARS-CoV-2: Percentage of participants with seroresponse

For the secondary immunogenicity endpoints, descriptive summaries statistics, including median, Q1, Q3, minimum, and maximum will be provided for each timepoints for the antibody titer values by treatment arm (available in Section 3.6.1) for the influenza and SARS-CoV-2 endpoints:

- GMT with corresponding 2-sided 95% CI
- GMFR of specific antibody titers with the corresponding 2-sided 95% CI at each post-basline timepoint Day 29 over pre-injection Baseline at Day 1

Additional descriptions will be provided by treatment arm (available in Section 3.6.1) for the following influenza and SARS-CoV-2 endpoints:

- Percentages of participants with seroconversion (influenza) and seroresponse (SARS-CoV-2) with the corresponding 2-sided 95% CI at each post-Baseline time point,
- Percentages of participants with a GMFR results >=2, and >=4 with the corresponding 2-sided 95% CI at each post-Baseline time point.

Reverse Cumulative Distribution Function for each specific strain of influenza and SARS-CoV-2 will be provided, as well as box plot and bar plot for GMT and GMFR, and bar plot for GMR, SCR and SRR at all evaluable timepoints.

# 3.6.4.3. Exploratory Immunogenicity Endpoints

The below exploratory analyses of immunogenicity may be performed:

- GMT and GMFR at all evaluable time points compared to Day 1 by HAI for influenza and PsVNA for SARS-CoV-2
- Influenza: Percentage of participants with seroconversion, as defined above
- SARS-CoV-2: Percentage of participants with seroresponse, as defined above

- GMT and GMFR at all evaluable time points compared to Day 1 by alternative methods, including, but not limited to: microneutralization assay for influenza or ligand-binding assay for SARS-CoV-2
- Frequency, specificities, or other endpoints to be determined for the further characterization of immune responses

# 3.6.5. Other Exploratory Endpoints

Transcriptomic and genomic samples will be part of the optional biomarker assessment. Exploratory assessments may include assessment of biomarkers for safety, reactogenicity, and inflammation. Serologic markers of disease severity, immune response to SARS-CoV-2 or influenza, reverse transcription polymerase chain reaction (RT-PCR) of nasal swab samples, genetic sequences of SARS-CoV-2 or influenza strains isolated from participants' samples, and genomic and transcriptomic samples may also be evaluated. Analyses and reporting of these endpoints will be covered in a separate analysis plan if applicable.

# 3.6.6. Planned Analyses

#### 3.6.6.1. Interim Analysis

An interim analysis of safety, reactogenicity, and immunogenicity is planned after all participants have completed the Day 29 visit. The interim analysis as of completion of Day 29 will be performed by the study statistician and programmers. The group-level unblinded summary data of the interim analyses may be reviewed by the Sponsor project team for safety monitoring and/or clinical development planning purposes for the mRNA-1083 project. More details will be documented in the study Data Blinding Plan.

# 3.6.6.2. Final Analysis

The final analysis will be performed after all participants in Part 2 have completed the Day 181/EoS visit.

# 4. Changes from Planned Analysis in Protocol

There are no changes in planned analysis.


#### 5. References

CDC, Centers for Disease Control and Prevention. 2020. Coronavirus Disease 2019 (COVID-19) 2020 Interim Case Definition, Approved August 5, 2020. [Online] August 2020. https://ndc.services.cdc.gov/case-definitions/coronavirus-disease-2019-2020-08-05/.

DHHS, Department of Health and Human Services, FDA, Food and Drug Administration, Center for Biologics Evaluation and Research (US). 2007. Guidance for industry: Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventative vaccine clinical trials. [Online] September 2007.

https://www.fda.gov/downloads/BiologicsBloodVaccines/GuidanceComplianceRegulatoryInformation/Guidances/Vaccines/ucm091977.pdf.

Nauta, Jozef. 2011. Statistics in Clinical Vaccine Trials. s.l.: Springer, 2011.

# 6. Appendices

# Appendix A Schedule of Activities (SoA)

# I. Part 1

| Visit Number | SCRN | 1 | 2 | 3 | 4, 5, 6, 7 | 8 | USV |
|---|---|---|---|---|---|---|---|
| Type of Visit | C | C | C | C | SC | C | C |
| Month Time Point | NA | | | M1 | M2-M5 | M6 | Up to M6 |
| Visit Day | SCRNa | D1<br>(Baseline) <sup>a</sup> | D8 | D29 | D57, D91,<br>D121,<br>D151 | D181/<br>EoS | NA |
| Window Allowance (Days) | -28 | NA | -1 to +3 | -7 to +3 | ±5 | ±14 | NA |
| Informed consent form,<br>demographics, concomitant<br>medications, medical history | X | | | | | | |
| Inclusion/exclusion criteria | X | X | | | | | |
| Blood collection for safety laboratory samples <sup>b</sup> | X | | X | | | | |
| Full physical examination <sup>c</sup> | X | | | | | | |
| Axillary lymph nodes assessment <sup>d</sup> | | X | | | | | |
| Symptom-directed physical examination <sup>e</sup> | | X | X | X | | X | X |
| Vital sign measurements <sup>f</sup> | X | X | | | | | |
| Electrocardiogram <sup>g</sup> | | X | | | | | |
| Pregnancy testing <sup>h</sup> | X | X | | | | | |
| Randomization | | X | | | | | |
| Study intervention (including 60-minute, postdose observation period) | | X | | | | | |
| Blood collection for humoral immunogenicity <sup>i</sup> | | X | | X | | X | |
| Blood collection for cellular immunogenicity <sup>i</sup> | | X | | X | | | |
| Optional blood collection for genomics <sup>j</sup> | | X | | | | | |
| Optional blood collection for transcriptomics <sup>j</sup> | | X | X | X | | | |
| Blood sample for potential cardiac biomarker analysis k | | X | | | | | |
| Nasal swab for virus detection <sup>l</sup> | | X | | | | | X |
| Blood collection for SARS-CoV-2 antibodies, nucleocapsid | | X | | | | | |
| eDiary activation for recording<br>solicited local and systemic ARs<br>(7 days) <sup>m</sup> | | X | | | | | |
| Review of solicited AR eDiary | | | X | | | | |
| Follow-up safety call <sup>n</sup> | | | | | X | | |

| Visit Number | SCRN | 1 | 2 | 3 | 4, 5, 6, 7 | 8 | USV |
|---|---|---|---|---|---|---|---|
| Type of Visit | С | С | C | C | SC | C | C |
| Month Time Point | NA | | | M1 | M2-M5 | M6 | Up to M6 |
| Visit Day | SCRNa | D1<br>(Baseline) <sup>a</sup> | D8 | D29 | D57, D91,<br>D121,<br>D151 | D181/<br>EoS | NA |
| Window Allowance (Days) | -28 | NA | -1 to +3 | -7 to +3 | ±5 | ±14 | NA |
| Recording of unsolicited AEs through Day 29 | | X | X | X | | | |
| Recording of SAEs, AESIs,<br>MAAEs, AEs leading to<br>discontinuation, and concomitant<br>medications associated with these<br>events | | X | X | X | X | X | X |
| Recording of nonstudy vaccinations | X | X | X | X | X | X | X |
| Study completion | | | | | | X | |

Abbreviations: AE=adverse event; AESI=adverse event of special interest; AR=adverse reaction;; C=clinic visit; COVID-19=coronavirus disease 2019; D=day; ECG=electrocardiogram; EoS=end of study; ILI=influenza-like illness; IM=intramuscular; M=month; MAAE=medically attended adverse event; NA=not applicable; - SAE=serious adverse event; SARS-CoV-2=severe acute respiratory syndrome coronavirus 2; SC=safety (telephone) call; SCRN=Screening; USV=unscheduled visit;

- a. Screening and Day 1 will NOT be performed on the same day. Additionally, the Screening Visit may be performed over multiple visits within the 28-day Screening window.
- b. Safety laboratory tests will consist of total white blood cell count, hemoglobin, hematocrit, platelets, aspartate aminotransferase, alanine aminotransferase, creatinine, alkaline phosphatase, and total bilirubin. Safety laboratory tests will be performed by the central laboratory.
- c. A full physical examination, including height and weight for calculation of body mass index, will be performed at Screening. Additional physical examinations may be performed during the study at the discretion of the Investigator.
- d. On the day of study intervention administration, prior to injection, axillary lymph nodes of the injection arm will be examined, and any abnormalities will be documented.
- e. Symptom-directed physical examinations will be performed at all clinic visits, except at Screening, where a full physical examination will be performed. Interim physical examinations will be performed at the discretion of the Investigator. Any clinically significant finding identified by a healthcare professional during postinjection study visits should be reported as an AE.
- f. Vital sign measurements: Systolic and diastolic blood pressure, heart rate, respiratory rate, and body temperature. The preferred route of temperature assessment is oral. Vital signs must be collected at Screening and on the day of injection (Day 1), once before and at least 60 minutes after injection. Vital signs may be collected at other clinic visits in conjunction with a symptom-directed physical examination. For all vital sign measurements, participant must be seated for 5 minutes before any measurements are
- g. For participants ≥18 to <51 years of age only: A 12-lead ECG will be obtained, after 10 minutes of supine rest, at Visit 1/Day 1 prior to injection. The purpose of the ECG is to serve as a stored Baseline comparison, should it be necessary, for subsequent clinical evaluation if a case of suspected myocarditis and/or pericarditis occurs within the conduct of the clinical trial. The ECG output should be filed in the participant's binder. Central reading of the ECG will not be performed. Incidental significant abnormal ECG findings should contribute to the Investigator's assessment of eligibility, at their discretion, as per Exclusion Criterion.
- h. For participants of childbearing potential, a point-of-care urine pregnancy test will be performed at the Screening Visit and before the IM injections on Day 1. At the discretion of the Investigator, a pregnancy test either via blood or point-of-care urine can be performed at any time. For participants of nonchildbearing potential, the follicle-stimulating hormone level may be measured at the Screening Visit, as necessary, and at the discretion of the Investigator, to confirm menopausal status.


ModernaTX, Inc. mRNA-1083-P101

- i. Baseline samples for humoral and cellular immunogenicity must be collected prior to receipt of injection on Day 1. Cellular immunogenicity will be sampled and assessed in a subset of participants.
- j. Transcriptomic and genomic samples will be part of the optional biomarker assessment once consented by the study participant. Blood draws on Day 1 must occur prior to participants being administered the study intervention.
- k. For participants ≥18 to <51 years of age only: Plasma and serum samples will be collected and banked for potential future cardiac biomarker assessment.
- 1. A nasal swab to test for the presence of viral respiratory pathogens will be collected prior to the study intervention administration on Day 1 to document any prevacination infection. A nasal swab should be collected through study completion for protocol-defined ILI or SARS-CoV-2 ≤7 days of symptom onset.
- m. The eDiary activiation and entries will be recorded by the participant starting approximately 60 minutes after injection while at the clinic with instruction provided by study staff. Study participants will continue to record in the eDiary each day after they leave the clinic, preferably in the evening and at the same time each day, on the day of injection and for 6 days following injection. Solicited local and systemic ARs will be recorded separately for each injection site.
- n. Trained study staff will call all participants to collect information related to any SAEs, MAAEs, AESIs, AEs leading to study discontinuation, information on concomitant medications associated with those events, and any nonstudy vaccinations.


## II. Part 2

| Visit Number | SCRN | 1 | 2 | 3 | 4, 5 | 6 | USV |
|---|---|---|---|---|---|---|---|
| Type of Visit | С | С | SC | C | SC | С | С |
| Month Timepoint | NA | | | M1 | M3-M5 | M6 | Up to M6 |
| Visit Day | SCRN <sup>a</sup> | D1<br>(Baseline) <sup>a</sup> | D8 | D29 | D91,<br>D151 | D181/<br>EoS | NA |
| Window Allowance (Days) | -28 | NA | -1 to +3 | -7 to +3 | ±5 | ±14 | NA |
| Informed consent form,<br>demographics, concomitant<br>medications, medical history | X | | | | | | |
| Inclusion/exclusion criteria | X | X | | | | | |
| Full physical examination <sup>b</sup> | X | | | | | | |
| Axillary lymph nodes assessment c | | X | | | | | |
| Symptom-directed physical examination <sup>d</sup> | | X | | X | | X | X |
| Vital sign measurements <sup>e</sup> | X | X | | | | | |
| Electrocardiogram f | | X | | | | | |
| Pregnancy testing <sup>g</sup> | X | X | | | | | |
| Randomization | | X | | | | | |
| Study intervention (including 60-minute, postdose observation period) | | X | | | | | |
| Blood collection for humoral immunogenicity h | | X | | X | | X | |
| Optional blood collection for genomics i | | X | | | | | |
| Optional blood collection for transcriptomics <sup>i</sup> | | X | | X | | | |
| Blood sample for potential cardiac biomarker analysis <sup>j</sup> | | X | | | | | |
| Nasal swab for virus detection k | | X | | | | | |
| Blood collection for SARS-CoV-2 antibodies, nucleocapsid | | X | | | | | |
| eDiary activation for recording solicited ARs (7 days) <sup>1</sup> | | X | | | | | |
| Review of solicited AR eDiary | | | X | | | | |
| Follow-up safety call m | | | X | | X | | |
| Recording of unsolicited AEs<br>through Day 29 | | X | X | X | | | |
| Recording of SAEs, AESIs,<br>MAAEs, AEs leading to<br>discontinuation, and concomitant<br>medications associated with these<br>events | | X | X | Х | Х | X | X |

| Visit Number | SCRN | 1 | 2 | 3 | 4, 5 | 6 | USV |
|---|---|---|---|---|---|---|---|
| Type of Visit | С | С | SC | C | SC | С | С |
| Month Timepoint | NA | | | M1 | M3-M5 | M6 | Up to M6 |
| Visit Day | SCRN <sup>a</sup> | D1<br>(Baseline) <sup>a</sup> | D8 | D29 | D91,<br>D151 | D181/<br>EoS | NA |
| Window Allowance (Days) | -28 | NA | -1 to +3 | -7 to +3 | ±5 | ±14 | NA |
| Recording of nonstudy vaccinations | X | X | X | X | X | X | X |
| Study completion | | | | | | X | |

Abbreviations: AE = adverse event; AESI = adverse event of special interest; AR = adverse reaction; BMI = body mass index; C = clinic visit; COVID-19 = coronavirus disease 2019; D = day; EoS = end of study; ILI = influenza-like illness; IM = intramuscular; M = month; MAAE = medically attended adverse event; NA = not applicable; SAE = serious adverse event; SARS-CoV-2 = severe acute respiratory syndrome coronavirus 2; SC = safety (telephone) call; SCRN = Screening; USV = unscheduled visit

- a. Screening and Day 1 may be performed on the same day or a different day. Additionally, the Screening Visit may be performed over multiple visits within the 28-day Screening window.
- b. A full physical examination, including height and weight for calculation of body mass index, will be performed at Screening. Additional physical examinations may be performed during the study at the discretion of the Investigator.
- c. On the day of study intervention administration, prior to injection, axillary lymph nodes of the injection arm will be examined, and any abnormalities will be documented.
- d. Symptom-directed physical examinations will be performed at all clinic visits, except at Screening, where a full physical examination will be performed. Interim physical examinations will be performed at the discretion of the Investigator. Any clinically significant finding identified by a healthcare professional during postinjection study visits should be reported as an AE.
- e. Vital sign measurements: Systolic and diastolic blood pressure, heart rate, respiratory rate, and body temperature. The preferred route of temperature assessment is oral. Vital signs must be collected at Screening and on the day of injection (Day 1), once before and at least 60 minutes after injection. Vital signs may be collected at other clinic visits in conjunction with a symptom-directed physical examination. For all vital sign measurements, participant must be seated for 5 minutes before any measurements are taken.
- f. A 12-lead ECG will be obtained, after 10 minutes of supine rest, at Visit 1/Day 1 prior to injection. The purpose of the ECG is to serve as a stored Baseline comparison, should it be necessary, for subsequent clinical evaluation if a case of suspected myocarditis and/or pericarditis occurs within the conduct of the clinical trial. The ECG output should be filed in the participant's binder. Central reading of the ECG will not be performed. Incidental significant abnormal ECG findings should contribute to the Investigator's assessment of eligibility, at their discretion, as per Exclusion Criterion.
- g. For participants of childbearing potential, a point-of-care urine pregnancy test will be performed at the Screening Visit and before the IM injections on Day 1. At the discretion of the Investigator, a pregnancy test either via blood or point-of-care urine can be performed at any time. For participants of nonchildbearing potential, the follicle-stimulating hormone level may be measured at the Screening Visit, as necessary, and at the discretion of the Investigator, to confirm menopausal status.
- h. Baseline samples for humoral immunogenicity must be collected prior to receipt of injection on Day 1.
- Transcriptomic and genomic samples will be part of the optional biomarker assessment once consented by the study participant. Blood draws on Day 1 must occur prior to participants being administered the study intervention.
- j. Plasma and serum samples will be collected prior to the study intervention administration on Day 1 and banked for potential future cardiac biomarker assessment.
- k. A nasal swab to test for the presence of viral respiratory pathogens will be collected prior to the study intervention administration on Day 1 to document any prevaccination infection.
- 1. The eDiary activation and entries will be recorded by the participant starting approximately 60 minutes after injection while at the clinic with instruction provided by study staff. Study participants will continue to record in the eDiary each day after they leave the clinic, preferably in the evening and at the same time each day, on


ModernaTX, Inc. mRNA-1083-P101

the day of injection and for 6 days following injection. Solicited local and systemic ARs will be recorded separately for each injection site.

m. Trained study staff will call all participants to collect information related to any SAEs, MAAEs, AESIs, AEs leading to study discontinuation, information on concomitant medications associated with those events, and any nonstudy vaccinations.


#### Appendix B Analysis Visit Windows

The following applies to Part 1 and Part 2:

Analysis visit windows will be utilized for immunogenicity assessments only.

Data will be mapped using the following approach:

Step 1: If the assessments are collected at a scheduled visit, the collected data will be mapped to the nominal scheduled visit.

Step 2: If the assessments are collected at an unscheduled visit, the collected data will be mapped using the analysis visit windows described in Table 16 below.

If a Participant has multiple assessments within the same analysis visit, the following rule will be used:

- If multiple assessments occur within a given analysis visit, the assessment closest to the target study day will be used.
- If there are 2 or more assessments equal distance to the target study day, the last assessment will be used.

**Table 16 Analysis Visit Windows for Immunogenicity Assessments** 

| Visit | Target Study Day | Visit Window in Study Day |
|---------|------------------|---------------------------|
| Day 1 | 1 | 1, Pre-vaccination |
| Day 29 | 29 | [2, 105] |
| Day 181 | 181 | ≥106 |

# Appendix C Imputation Rules for Missing Prior/Concomitant Medications and Non-Study Vaccinations

The following applies to Part 1 and Part 2:

Imputation rules for missing or partial medication start/stop dates are defined below:

- a) Missing or partially missing medication start date:
  - If only Day is missing, use the first day of the month, unless the start month and year of the medication coincide with the start month and year of the IP injection.
    - If not marked as a prior medication on the Prior/Concomitant CRF page ("Was
      the medication taken prior to study administration?" = "No"), then use the date of
      the IP injection.
    - If marked as a prior medication on the Prior/Concomitant CRF page ("Was the medication taken prior to study administration?" = "Yes"), then use the earlier of the first day of the month or the date of the IP injection 1.
    - If the mark on the Prior/Concomitant CRF page ("Was the medication taken prior to study administration?") is missing and the medication end date is on/after the date of the IP injection or is missing, then use the date of the IP injection.
  - If Day and Month are both missing, use the first day of the year, unless the start year of the medication coincide with the start year of the IP injection.
    - If not marked as a prior medication on the Prior/Concomitant CRF page ("Was
      the medication taken prior to study administration?" = "No"), then use the date of
      the IP injection.
    - If marked as a prior medication on the Prior/Concomitant CRF page ("Was the medication taken prior to study administration?" = "Yes"), then use the earlier of the first day of the year or the date of the IP injection -1.
    - If the mark on the Prior/Concomitant CRF page ("Was the medication taken prior to study administration?") is missing and the medication end date is on/after the date of the IP injection or is missing, then use the date of the IP injection.
  - If Day, Month and Year are all missing, the date will not be imputed, but will use the following rules for purposes of determining the status as prior and/or concomitant.
    - If not marked as a prior medication on the Prior/Concomitant CRF page ("Was
      the medication taken prior to study administration?" = "No"), then the medication
      will be treated as having begun after IP injection.
    - If marked as a prior medication on the Prior/Concomitant CRF page ("Was the medication taken prior to study administration?" = "Yes"), or if the mark is missing, then the medication will be treated as a prior medication (and as a concomitant medication unless the stop date indicates the medication was stopped prior to IP injection).
- b) Missing or partial medication stop date:

- If only Day is missing, use the earliest date of (last day of the month, study completion, discontinuation from the study, or death).
- If Day and Month are both missing, use the earliest date of (last day of the year, study completion, discontinuation from the study, or death).
- If Day, Month and Year are all missing, the date will not be imputed, but the medication will be flagged as a continuing medication.

In summary, the prior, concomitant or post categorization of a medication is described in Table 17 below.

Table 17 Prior, Concomitant, and Post Categorization of a Medication

| | <b>Medication Stop Date</b> | | |
|---|---|---|---|
| Medication Start Date | < Injection Date | ≥ Injection Date and ≤<br>Injection Date + 27<br>days | > 27 Days After<br>Injection [2] |
| < Injection Date [1] | P | PC | PCA |
| $\geq$ Injection date and $\leq$ 27 days after injection | - | C | CA |
| > 27 days after injection | - | - | A |

A: Post; C: Concomitant; P: Prior

- [1] includes medications with completely missing start date
- [2] includes medications with completely missing end date

#### **Appendix D** Imputation Rules for Missing AE dates

The following applies to Part 1 and Part 2:

Imputation rules for missing or partial AE start dates and stop dates are defined below:

- a) Missing or partial AE start date:
  - If only DAY is missing, use the first day of the month, unless:
    - The AE end date is after the date of injection or is missing AND the start month and year of the AE coincide with the start month and year of the injection. In this case, use the date and time of injection, even if time is collected.
  - If DAY and Month are both missing, use the first day of the year, unless:
    - The AE end date is after the date of injection or is missing AND the start year of the AE coincides with the start year of the injection. In this case, use the date of injection
  - If DAY, Month and Year are all missing, the date will not be imputed. However, if the AE end date is prior to the date of injection, then the AE will be considered a pretreatment AE. Otherwise, the AE will be considered treatment emergent.
- b) Missing or partial AE end dates will not be imputed.


#### **Appendix E** Severity Grading of Laboratory Abnormalities

The following applies to Part 1 only:

| Serum* | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4)** |
|---|---|---|---|---|
| Sodium – Hyponatremia mEq/L | 132 - 134 | 130 – 131 | 125 – 129 | < 125 |
| Sodium – Hypernatremia mEq/L | 144 - 145 | 146 – 147 | 148 – 150 | > 150 |
| Potassium – Hyperkalemia mEq/L | 5.1 - 5.2 | 5.3 - 5.4 | 5.5 - 5.6 | > 5.6 |
| Potassium – Hypokalemia mEq/L | 3.5 - 3.6 | 3.3 - 3.4 | 3.1 - 3.2 | < 3.1 |
| Glucose – Hypoglycemia mg/dL | 65 – 69 | 55 – 64 | 45 – 54 | < 45 |
| Glucose – Hyperglycemia<br>Fasting – mg/dL<br>Random – mg/dL | 100 – 110<br>110 – 125 | 111 – 125<br>126 – 200 | >125<br>>200 | Insulin requirements or hyperosmolar coma |
| Blood Urea Nitrogen (BUN) mg/dL | 23 - 26 | 27 - 31 | > 31 | Requires dialysis |
| Creatinine – mg/dL | 1.5 – 1.7 | 1.8 - 2.0 | 2.1 – 2.5 | > 2.5 or requires dialysis |
| Calcium – hypocalcemia mg/dL | 8.0 - 8.4 | 7.5 - 7.9 | 7.0 - 7.4 | < 7.0 |
| Calcium – hypercalcemia mg/dL | 10.5 - 11.0 | 11.1 – 11.5 | 11.6 - 12.0 | > 12.0 |
| Magnesium – hypomagnesemia mg/dL | 1.3 – 1.5 | 1.1 – 1.2 | 0.9 – 1.0 | < 0.9 |
| Phosphorous – hypophosphatemia mg/dL | 2.3 - 2.5 | 2.0 - 2.2 | 1.6 – 1.9 | < 1.6 |
| CPK – mg/dL | 1.25 – 1.5 x<br>ULN*** | 1.6 – 3.0 x ULN | 3.1 – 10 x ULN | > 10 x ULN |
| Albumin – Hypoalbuminemia g/dL | 2.8 - 3.1 | 2.5 - 2.7 | < 2.5 | |
| Total Protein – Hypoproteinemia g/dL | 5.5 – 6.0 | 5.0 – 5.4 | < 5.0 | |
| Alkaline phosphate – increase by factor | 1.1 – 2.0 x<br>ULN | 2.1 – 3.0 x ULN | 3.1 – 10 x ULN | > 10 x ULN |
| Liver Function Tests –ALT, AST increase by factor | 1.1 – 2.5 x<br>ULN | 2.6 – 5.0 x ULN | 5.1 – 10 x ULN | > 10 x ULN |
| Bilirubin – when accompanied by<br>any increase in Liver Function Test<br>increase by factor | 1.1 – 1.25 x<br>ULN | 1.26 – 1.5 x<br>ULN | 1.51 – 1.75 x<br>ULN | > 1.75 x ULN |
| Bilirubin – when Liver Function<br>Test is normal; increase by factor | 1.1 – 1.5 x<br>ULN | 1.6 – 2.0 x ULN | 2.0 - 3.0 x ULN | > 3.0 x ULN |
| Cholesterol | 201 – 210 | 211 – 225 | > 226 | |
| Pancreatic enzymes – amylase, lipase | 1.1 – 1.5 x<br>ULN | 1.6 – 2.0 x ULN | 2.1 – 5.0 x ULN | > 5.0 x ULN |

<sup>\*</sup> The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.


<sup>\*\*</sup> The clinical signs or symptoms associated with laboratory abnormalities might result in characterization of the laboratory abnormalities as Potentially Life Threatening (Grade 4). For example. A low sodium value that falls within a Grade 3 parameter (125-129 mE/L) should be recorded as a Grade 4 hyponatremia event if the participant had a new seizure associated with the low sodium value.

<sup>\*\*\*</sup>ULN" is the upper limit of the normal range.

| Hematology * | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening (Grade<br>4) |
|---|---|---|---|---|
| Hemoglobin (Female) – mg/dL | 11.0 – 12.0 | 9.5 – 10.9 | 8.0 – 9.4 | < 8.0 |
| Hemoglobin (Female)<br>change from baseline<br>value – mg/dL | Any decrease – 1.5 | 1.6 – 2.0 | 2.1 – 5.0 | > 5.0 |
| Hemoglobin (Male) – mg/dL | 12.5 – 13.5 | 10.5 – 12.4 | 8.5 – 10.4 | < 8.5 |
| Hemoglobin (Male)<br>change from baseline<br>value – mg/dL | Any decrease – 1.5 | 1.6 – 2.0 | 2.1 – 5.0 | > 5.0 |
| WBC Increase – cell/mm <sup>3</sup> | 10,800 - 15,000 | 15,001 - 20,000 | 20,001 - 25,000 | > 25,000 |
| WBC Decrease – cell/mm <sup>3</sup> | 2,500 - 3,500 | 1,500 - 2,499 | 1,000 - 1,499 | < 1,000 |
| Lymphocytes Decrease – cell/mm <sup>3</sup> | 750 – 1,000 | 500 – 749 | 250 – 499 | < 250 |
| Neutrophils Decrease – cell/mm <sup>3</sup> | 1,500 – 2,000 | 1,000 – 1,499 | 500 – 999 | < 500 |
| Eosinophils – cell/mm <sup>3</sup> | 650 - 1500 | 1501 - 5000 | > 5000 | Hypereosinophilic |
| Platelets Decreased – cell/mm <sup>3</sup> | 125,000 –<br>140,000 | 100,000 –<br>124,000 | 25,000 – 99,000 | < 25,000 |
| PT – increase by factor (prothrombin time) | 1.0 – 1.10 x<br>ULN** | 1.11 – 1.20 x<br>ULN | 1.21 – 1.25 x<br>ULN | > 1.25 ULN |
| PTT – increase by factor (partial thromboplastin time) | 1.0 – 1.2 x ULN | 1.21 – 1.4 x ULN | 1.41 – 1.5 x ULN | > 1.5 x ULN |
| Fibrinogen increase – mg/dL | 400 – 500 | 501 – 600 | > 600 | |
| Fibrinogen decrease – mg/dL | 150 – 200 | 125 – 149 | 100 – 124 | < 100 or associated<br>with gross bleeding<br>or disseminated<br>intravascular<br>coagulation (DIC) |

<sup>\*</sup> The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.

\*\* "ULN" is the upper limit of the normal range.

## **Appendix F** Severity Grading of Vital Sign Abnormalities

The following applies to Part 1 and Part 2:

| Vital Signs* | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Fever (°C)**<br>(°F)** | 38.0 – 38.4<br>100.4 – 101.1 | 38.5 - 38.9 $101.2 - 102.0$ | 39.0 – 40<br>102.1 – 104 | > 40<br>> 104 |
| Tachycardia - beats per minute | 101 – 115 | 116 – 130 | > 130 | ER visit or<br>hospitalization for<br>arrhythmia |
| Bradycardia - beats per minute*** | 50 – 54 | 45 – 49 | < 45 | ER visit or<br>hospitalization for<br>arrhythmia |
| Hypertension (systolic) - mm<br>Hg | 141 – 150 | 151 – 155 | > 155 | ER visit or<br>hospitalization for<br>malignant hypertension |
| Hypertension (diastolic) -<br>mm Hg | 91 – 95 | 96 – 100 | > 100 | ER visit or hospitalization for malignant hypertension |
| Hypotension (systolic) – mm<br>Hg | 85 – 89 | 80 – 84 | < 80 | ER visit or<br>hospitalization for<br>hypotensive shock |
| Respiratory Rate – breaths per minute | 17 – 20 | 21 – 25 | > 25 | Intubation |

<sup>\*</sup> Participant should be at rest for all vital sign measurements.

<sup>\*\*</sup> Oral temperature; no recent hot or cold beverages or smoking.

<sup>\*\*\*</sup> When resting heart rate is between 60 – 100 beats per minute. Use clinical judgement when characterizing bradycardia among some healthy participant populations, for example, conditioned athletes.

# **Appendix G** Solicited Adverse Reactions and Grades

The following applies to Part 1 and Part 2:

| Reaction | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|---|
| Injection site pain | None | | | Prevents daily activity | Requires<br>emergency room<br>visit or<br>hospitalization |
| Injection site erythema (redness) | <25 mm/<br><2.5 cm | 25 to 50 mm/<br>2.5 to 5 cm | 51 to 100 mm/<br>5.1 to 10 cm | >100 mm/<br>>10 cm | Necrosis or exfoliative dermatitis |
| Injection site<br>swelling/ induration<br>(hardness) | <25 mm/<br><2.5 cm | 25 to 50 mm/<br>2.5 to 5 cm | 51 to 100 mm/<br>5.1 to 10 cm | >100 mm/<br>>10 cm | Necrosis |
| Axillary (underarm) swelling or tenderness ipsilateral to the side of injection | None | No interference with activity | Some interference with activity | Prevents daily activity | Emergency<br>room visit or<br>hospitalization |
| Headache | None | No interference with activity | Some interference with activity | Prevents daily activity | Requires<br>emergency room<br>visit or<br>hospitalization |
| Fatigue | None | No interference with activity | Some interference with activity | Prevents daily activity | Requires<br>emergency room<br>visit or<br>hospitalization |
| Myalgia (muscle<br>aches all over body) | None | No interference with activity | Some interference with activity | Prevents daily activity | Requires<br>emergency room<br>visit or<br>hospitalization |
| Arthralgia (joint aches in several joints) | None | No interference with activity | Some interference with activity | Prevents daily activity | Requires<br>emergency room<br>visit or<br>hospitalization |
| Nausea/vomiting | None | No interference<br>with activity or 1<br>to 2 episodes/<br>24 hours | Some interference with activity or >2 episodes/ 24 hours | Prevents daily<br>activity, requires<br>outpatient<br>intravenous<br>hydration | Requires<br>emergency room<br>visit or<br>hospitalization<br>for hypotensive<br>shock |

| Reaction | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|---|
| Chills | None | No interference with activity | Some interference with activity not requiring medical intervention | Prevents daily<br>activity and<br>requires medical<br>intervention | Requires<br>emergency room<br>visit or<br>hospitalization |
| Fever (oral) | <38.0°C<br><100.4°F | 38.0 to 38.4°C<br>100.4 to 101.1°F | 38.5 to 38.9°C<br>101.2 to 102.0°F | 39.0 to 40.0°C<br>102.1 to 104.0°F | >40.0°C<br>>104.0°F |

Note: Events listed above but starting >7 days post study intervention administration will be recorded on the AE page of the electronic case report form (eCRF). Causality for each event will be determined per assessment by the Investigator.


# Appendix H TEAE of Specifical Interest by SMQ

The following applies to Part 1 and Part 2:

| SMQ/CMQ Name* | Type of<br>MedDRA<br>Query | SMQ<br>Level | SMQ Code | Broad or Narrow<br>Search |
|---|---|---|---|---|
| Anaphylactic Reaction | SMQ | 1 | 20000021 | Algorithm |
| | | | | A or (B and C) or (D and (B or C)) |
| Angioedema | SMQ | 1 | 20000024 | Narrow |
| Arthritis | SMQ | 1 | 20000216 | Narrow |
| Cardiac Arrhythmias | SMQ | 1 | 20000049 | Narrow |
| Arrhythmia Related Investigations, Signs and Symptoms | SMQ | 2 | 20000051 | Narrow |
| Cardiac Arrhythmia Terms (including bradyarrhythmias and tachyarrhythmias) | SMQ | 2 | 20000050 | Narrow |
| Cardiac Failure | SMQ | 1 | 20000004 | Narrow |
| Cardiomyopathy | SMQ | 1 | 20000150 | Narrow |
| Central Nervous System Vascular Disorders | SMQ | 1 | 20000060 | Narrow |
| Central Nervous System Haemorrhages and<br>Cerebrovascular Conditions | SMQ | 2 | 20000061 | Narrow |
| Central Nervous System Vascular Disorders, not<br>Specified as Haemorrhagic or Ischaemic | SMQ | 2 | 20000165 | Narrow |
| Convulsions | SMQ | 1 | 20000079 | Narrow |
| Demyelination | SMQ | 1 | 20000154 | Narrow |
| Embolic and Thrombotic Events | SMQ | 1 | 20000081 | Narrow |
| Embolic and Thrombotic Events, Arterial | SMQ | 2 | 20000082 | Narrow |
| Embolic and Thrombotic Events, Venous | SMQ | 2 | 20000084 | Narrow |
| Embolic and Thrombotic Events, Vessel Type<br>Unspecified and Mixed Arterial and Venous | SMQ | 2 | 20000083 | Narrow |
| Guillain-Barre Syndrome | SMQ | 1 | 20000131 | Narrow |
| Haematopoietic Cytopenias | SMQ | 1 | 20000027 | Narrow |
| Haematopoietic Cytopenias Affecting More Than<br>One Type Of Blood Cell | SMQ | 2 | 20000028 | Narrow |
| Haematopoietic Erythropenia | SMQ | 2 | 20000029 | Narrow |
| Haematopoietic Leukopenia | SMQ | 2 | 20000030 | Narrow |
| Haematopoietic Thrombocytopenia | SMQ | 2 | 20000031 | Narrow |
| Hearing and Vestibular Disorders | SMQ | 1 | 20000170 | Narrow |
| Hearing Impairment | SMQ | 2 | 20000171 | Narrow |
| Vestibular Disorders | SMQ | 2 | 20000172 | Narrow |
| Hypersensitivity | SMQ | 1 | 20000214 | Narrow |
| Immune-mediated/Autoimmune Disorders | SMQ | 1 | 20000236 | Narrow |
| Ischaemic Heart Disease | SMQ | 1 | 20000043 | Narrow |
| Myocardial Infarction | SMQ | 2 | 20000047 | Narrow |

| Other Ischaemic Heart Disease | SMQ | 2 | 20000168 | Narrow |
|----------------------------------------|-----|---|----------|--------|
| Noninfectious Myocarditis/Pericarditis | SMQ | 1 | 20000239 | Narrow |
| Peripheral Neuropathy | SMQ | 1 | 20000034 | Narrow |
| Thrombophlebitis | SMQ | 1 | 20000115 | Narrow |
| Vasculitis | SMQ | 1 | 20000174 | Narrow |

<sup>\*</sup> Based on MedDRA 26.1

#### Algorithmic Approach for Anaphylactic Reaction:

The following criteria will be used to determine anaphylactic reaction:

- a) A term from Category A or
- b) A term from Category B (Upper Airway/Respiratory) and a term from Category C (Angioedema/Urticaria/Pruritus/Flush) that occurred within 24 hours of each other or
- c) A term from Category D (Cardiovascular/Hypotension) and at least one of the following:
  - A term from Category B (Upper Airway/Respiratory) that occurred within 24 hours of each other.
  - A term from Category C (Angioedema/Urticaria/Pruritus/Flush) that occurred within 24 hours of each other.

| Anaphylactic Reaction | | |
|---|---|---|
| Category | ory Scope PT Search Term | |
| A | Narrow | Anaphylactic reaction |
| A | Narrow | Anaphylactic shock |
| A | Narrow | Anaphylactic transfusion reaction |
| A | Narrow | Anaphylactoid reaction |
| A | Narrow | Anaphylactoid shock |
| A | Narrow | Circulatory collapse |
| A | Narrow | Dialysis membrane reaction |
| A | Narrow | Kounis syndrome |
| A | Narrow | Procedural shock |
| A | Narrow | Shock |
| A | Narrow | Shock symptom |
| A | Narrow | Type I hypersensitivity |
| В | Broad | Asthma |
| В | Broad | Bronchial oedema |
| В | Broad | Bronchospasm |
| В | Broad | Cardio-respiratory distress |
| В | Broad | Chest discomfort |
| В | Broad | Choking |
| В | Broad | Choking sensation |
| В | Broad | Circumoral oedema |

| Anaphylactic Reaction | | |
|---|---|---|
| Category | Scope | PT Search Term |
| В | Broad | Cough |
| В | Broad | Cough variant asthma |
| В | Broad | Cyanosis |
| В | Broad | Dyspnoea |
| В | Broad | Enhanced respiratory disease |
| В | Broad | Hyperventilation |
| В | Broad | Irregular breathing |
| В | Broad | Laryngeal dyspnoea |
| В | Broad | Laryngeal oedema |
| В | Broad | Laryngospasm |
| В | Broad | Laryngotracheal oedema |
| В | Broad | Mouth swelling |
| В | Broad | Nasal obstruction |
| В | Broad | Oedema mouth |
| В | Broad | Oropharyngeal oedema |
| В | Broad | Oropharyngeal spasm |
| В | Broad | Oropharyngeal swelling |
| В | Broad | Pharyngeal oedema |
| В | Broad | Pharyngeal swelling |
| В | Broad | Respiratory arrest |
| В | Broad | Respiratory distress |
| В | Broad | Respiratory failure |
| В | Broad | Reversible airways obstruction |
| В | Broad | Sensation of foreign body |
| В | Broad | Sneezing |
| В | Broad | Stridor |
| В | Broad | Swollen tongue |
| В | Broad | Tachypnoea |
| В | Broad | Throat tightness |
| В | Broad | Tongue oedema |
| В | Broad | Tracheal obstruction |
| В | Broad | Tracheal oedema |
| В | Broad | Upper airway obstruction |
| В | Broad | Vaccine associated enhanced respiratory disease |
| В | Broad | Wheezing |
| C | Broad | Allergic oedema |
| С | Broad | Angioedema |
| C | Broad | Circumoral swelling |
| C | Broad | Erythema |
| C | Broad | Eye oedema |
| C | Broad | Eye pruritus |
| C | Broad | Eye swelling |
| C | Broad | Eyelid oedema |
| C | Broad | Face oedema |
| C | Broad | Flushing |
| C | Broad | Injection site urticaria |
| C | Broad | Lip oedema |
| C | Broad | Lip swelling |
| C | Broad | Nodular rash |
| C | Broad | Ocular hyperaemia |
| | DIVIU | Could 13 perueiniu |

| Anaphylactic Reaction | | |
|-----------------------|-------|------------------------------------|
| Category | Scope | PT Search Term |
| С | Broad | Oedema |
| С | Broad | Oedema blister |
| С | Broad | Periorbital oedema |
| С | Broad | Periorbital swelling |
| С | Broad | Pruritus |
| С | Broad | Pruritus allergic |
| С | Broad | Rash |
| C | Broad | Rash erythematous |
| C | Broad | Rash pruritic |
| С | Broad | Skin swelling |
| С | Broad | Swelling |
| С | Broad | Swelling face |
| С | Broad | Swelling of eyelid |
| С | Broad | Urticaria |
| С | Broad | Urticaria papular |
| D | Broad | Blood pressure decreased |
| D | Broad | Blood pressure diastolic decreased |
| D | Broad | Blood pressure systolic decreased |
| D | Broad | Cardiac arrest |
| D | Broad | Cardio-respiratory arrest |
| D | Broad | Cardiovascular insufficiency |
| D | Broad | Diastolic hypotension |
| D | Broad | Hypotension |
| D | Broad | Hypotensive crisis |
| D | Broad | Post procedural hypotension |